CLINICAL TRIAL: NCT01126437
Title: A Randomized, Active-controlled, Double-blind, Double-dummy, Parallel Group Design, Multi-center Trial to Compare the Efficacy and Safety of 2.5 µg and 5 µg Tiotropium Inhalation Solution Delivered by the Respimat Inhaler With Tiotropium Inhalation Capsules 18 µg Delivered by the HandiHaler (TIOSPIR)
Brief Title: Comparison of Tiotropium in the HandiHaler Versus the Respimat in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.452; 2009-015713-51 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-05-06; First posted 2010-05-19 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

ARMS (3):
- tiotropium 2.5 mcg and placebo (Experimental): Patients receive one of the active tiotropium arms daily
  Interventions: Drug: tiotropium 1.25 mcg (2 actuations/day)
- tiotropium 18 mcg and placebo (Active Comparator): Patients receive one of the active tiotropium arms daily
  Interventions: Drug: tiotropium 18 mcg
- tiotropium 5 mcg and placebo (Experimental): Patients receive one of the active tiotropium arms daily
  Interventions: Drug: tiotropium 2.5 mcg (2 actuations/day)

INTERVENTIONS:
Drug: tiotropium 18 mcg — HandiHaler
  Arms: tiotropium 18 mcg and placebo
Drug: tiotropium 1.25 mcg (2 actuations/day) — soft mist inhaler 2 actuations=2 puffs/day
  Arms: tiotropium 2.5 mcg and placebo
Drug: tiotropium 2.5 mcg (2 actuations/day) — soft mist inhaler (2 actuations=2 puffs/day)
  Arms: tiotropium 5 mcg and placebo

SUMMARY:
Direct comparison studies of the tiotropium HandiHaler® 18 µg and Respimat® 5 µg formulations have been limited to 4-week crossover studies. Therefore, prospective data from a trial of adequate size and duration is required to establish that compared to tiotropium HandiHaler®, tiotropium Respimat® will have (a) similar effects on safety and (b) similar or superior effects on exacerbations.

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign an informed consent consistent with International Conference on Harmonization Good Clinical Practice (ICH-GCP) guidelines prior to participation in the trial, which includes medication washout and restrictions.
2. Male or female patients 40 years of age or older.
3. Patients must be current or ex-smokers with a smoking history of ≥10 pack-years. (Patients who have never smoked cigarettes must be excluded)
4. All patients must have a diagnosis of COPD (P06-12085), and must meet the following criteria: Relatively stable airway obstruction with a post-bronchodilator FEV1 ≤ 70% of predicted normal and post-bronchodilator FEV1 / FVC ≤70%.

   Pulmonary function tests (PFTs) were conducted after the inhalation of 400 μg salbutamol / albuterol (preferred), however testing with either 200 μg salbutamol/albuterol or a combination of salbutamol / albuterol with ipratropium bromide (2 to 4 actuations) was acceptable. Other short-acting beta agonists, such as terbutaline, may have been used for the testing. The medication used for the testing was documented. Further, historical data from measurements within the past 6 months either at the site or at a referral site may have been used (see Section 6.2.1 of the CTP, located in Appendix 16.1.1). Subjects were not to have been randomized to the study without the availability of spirometry data at the actual study site.

   Eligibility for PFT sub-study: For subjects participating in the spirometry sub-study, historical data may not have been used for inclusion. These subjects must have qualified in the clinic at Visit 1 after performing a baseline measurement. These subjects performed a pre-dose PFT which was followed by the administration of 400 μg salbutamol / albuterol only (no other short-acting beta agonist was allowed), followed by a post-dose PFT for qualification.
5. Able to inhale from the HandiHaler® and the Respimat® devices.

Exclusion criteria:

1. Significant diseases other than COPD. A significant disease is defined as a disease or condition which, in the opinion of the investigator, may put the patient at risk because of participation in the study or may influence the patients ability to participate in the study.
2. Patients with a recent history (i.e., six months or less) of myocardial infarction.
3. Patients with any unstable or life-threatening cardiac arrhythmia requiring intervention or change in drug therapy during the last year.
4. Hospitalisation for cardiac failure (New York Heart Association (NYHA) Class III or IV) during the past year.
5. Known active tuberculosis.
6. Patients with a history of asthma, cystic fibrosis, clinically evident bronchiectasis, interstitial lung disease, or pulmonary thromboembolic disease.
7. History of thoracotomy with pulmonary resection. Subjects with a history of thoracotomy for other reasons were to have been evaluated per exclusion criterion 1.
8. Subject was planning to undergo lung transplant or lung volume reduction surgery (LVRS).
9. Malignancy for which the subject had undergone resection, radiation, chemotherapy or biological treatments within the last 5 years. Subjects with treated basal cell carcinoma were allowed.
10. Known respiratory infection or exacerbation of COPD in the 4 weeks prior to randomization.
11. Known hypersensitivity to anticholinergic drugs, lactose, benzalkonium chloride (BAC), ethylenediaminetetraacetic acid (EDTA), or any other components of the HandiHaler® or Respimat® inhalation solution delivery system.
12. Known moderate to severe renal impairment (as judged by the investigator).
13. Known narrow angle glaucoma.
14. Known significant symptomatic prostatic hyperplasia or bladder-neck obstruction. Subjects whose symptoms were controlled on treatment may have been included.
15. Use of systemic corticosteroid medication at unstable doses (i.e., less than 6 weeks on stable dose) or at doses in excess of the equivalent of 10 mg prednisolone per day.
16. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception for at least 3 months prior to and for the duration of the trial.
17. Significant alcohol or drug abuse within the past 12 months.
18. Subjects requiring the use of supplemental oxygen therapy for > 12 hours per day.
19. Subjects who had completed a pulmonary rehabilitation program in the 6 weeks prior to the screening visit or subjects who were currently in a pulmonary rehabilitation program that was not maintained throughout the duration of the study.
20. Subjects who had taken an investigational drug within 30 days prior to the Screening Visit.
21. Previous participation (receipt of randomized treatment) in this study.
22. Subjects who were currently participating in an interventional study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17183 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1191):
- United States (303):
  - 205.452.01107 Boehringer Ingelheim Investigational Site, Athens, Alabama
  - 205.452.01023 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 205.452.01035 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 205.452.01052 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 205.452.01219 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 205.452.01227 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 205.452.01280 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 205.452.01198 Boehringer Ingelheim Investigational Site, Florence, Alabama
  - 205.452.01244 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 205.452.01041 Boehringer Ingelheim Investigational Site, Montgomery, Alabama
  - 205.452.01070 Boehringer Ingelheim Investigational Site, Anchorage, Alaska
  - 205.452.01218 Boehringer Ingelheim Investigational Site, Chandler, Arizona
  - 205.452.01175 Boehringer Ingelheim Investigational Site, Mesa, Arizona
  - 205.452.01200 Boehringer Ingelheim Investigational Site, Mesa, Arizona
  - 205.452.01317 Boehringer Ingelheim Investigational Site, Mesa, Arizona
  - 205.452.01350 Boehringer Ingelheim Investigational Site, Pheonix, Arizona
  - 205.452.01254 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 205.452.01283 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 205.452.01315 Boehringer Ingelheim Investigational Site, Tempe, Arizona
  - 205.452.01158 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 205.452.01161 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 205.452.01302 Boehringer Ingelheim Investigational Site, Anaheim, California
  - 205.452.01038 Boehringer Ingelheim Investigational Site, Encinitas, California
  - 205.452.01313 Boehringer Ingelheim Investigational Site, Fountain Valley, California
  - 205.452.01375 Boehringer Ingelheim Investigational Site, Fountain Valley, California
  - 205.452.01074 Boehringer Ingelheim Investigational Site, Fullerton, California
  - 205.452.01345 Boehringer Ingelheim Investigational Site, Lancaster, California
  - 205.452.01171 Boehringer Ingelheim Investigational Site, Lincoln, California
  - 205.452.01339 Boehringer Ingelheim Investigational Site, Lomita, California
  - 205.452.01298 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 205.452.01356 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 205.452.01148 Boehringer Ingelheim Investigational Site, Orange, California
  - 205.452.01111 Boehringer Ingelheim Investigational Site, Palm Springs, California
  - 205.452.01147 Boehringer Ingelheim Investigational Site, Paramount, California
  - 205.452.01071 Boehringer Ingelheim Investigational Site, Poway, California
  - 205.452.01089 Boehringer Ingelheim Investigational Site, Rancho Cucamonga, California
  - 205.452.01097 Boehringer Ingelheim Investigational Site, Redlands, California
  - 205.452.01078 Boehringer Ingelheim Investigational Site, San Diego, California
  - 205.452.01176 Boehringer Ingelheim Investigational Site, San Diego, California
  - 205.452.01346 Boehringer Ingelheim Investigational Site, San Diego, California
  - 205.452.01306 Boehringer Ingelheim Investigational Site, San Jose, California
  - 205.452.01297 Boehringer Ingelheim Investigational Site, Santa Barbara, California
  - 205.452.01362 Boehringer Ingelheim Investigational Site, Tustin, California
  - 205.452.01225 Boehringer Ingelheim Investigational Site, Victorville, California
  - 205.452.01224 Boehringer Ingelheim Investigational Site, Walnut Creek, California
  - 205.452.01236 Boehringer Ingelheim Investigational Site, Wildomar, California
  - 205.452.01049 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 205.452.01245 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 205.452.01351 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 205.452.01018 Boehringer Ingelheim Investigational Site, Fort Collins, Colorado
  - 205.452.01005 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 205.452.01024 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 205.452.01199 Boehringer Ingelheim Investigational Site, Danbury, Connecticut
  - 205.452.01054 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 205.452.01072 Boehringer Ingelheim Investigational Site, Norwalk, Connecticut
  - 205.452.01040 Boehringer Ingelheim Investigational Site, Stamford, Connecticut
  - 205.452.01109 Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - 205.452.01308 Boehringer Ingelheim Investigational Site, Newark, Delaware
  - 205.452.01011 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 205.452.01209 Boehringer Ingelheim Investigational Site, Hialeah, Florida
  - 205.452.01360 Boehringer Ingelheim Investigational Site, Homestead, Florida
  - 205.452.01241 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 205.452.01337 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 205.452.01343 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 205.452.01184 Boehringer Ingelheim Investigational Site, Jupiter, Florida
  - 205.452.01138 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 205.452.01246 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 205.452.01321 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 205.452.01290 Boehringer Ingelheim Investigational Site, New Port Richey, Florida
  - 205.452.01203 Boehringer Ingelheim Investigational Site, Ocala, Florida
  - 205.452.01174 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 205.452.01135 Boehringer Ingelheim Investigational Site, Ormond Beach, Florida
  - 205.452.01173 Boehringer Ingelheim Investigational Site, Oviedo, Florida
  - 205.452.01195 Boehringer Ingelheim Investigational Site, Panama City, Florida
  - 205.452.01197 Boehringer Ingelheim Investigational Site, Panama City, Florida
  - 205.452.01239 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 205.452.01247 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 205.452.01286 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 205.452.01240 Boehringer Ingelheim Investigational Site, Pensacola, Florida
  - 205.452.01260 Boehringer Ingelheim Investigational Site, Ponte Vedra, Florida
  - 205.452.01092 Boehringer Ingelheim Investigational Site, Rockledge, Florida
  - 205.452.01251 Boehringer Ingelheim Investigational Site, Sarasota, Florida
  - 205.452.01133 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 205.452.01136 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 205.452.01207 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 205.452.01134 Boehringer Ingelheim Investigational Site, Tamarac, Florida
  - 205.452.01231 Boehringer Ingelheim Investigational Site, Tamarac, Florida
  - 205.452.01025 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 205.452.01250 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 205.452.01060 Boehringer Ingelheim Investigational Site, Winter Park, Florida
  - 205.452.01130 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 205.452.01047 Boehringer Ingelheim Investigational Site, Austell, Georgia
  - 205.452.01255 Boehringer Ingelheim Investigational Site, Columbus, Georgia
  - 205.452.01012 Boehringer Ingelheim Investigational Site, Conyers, Georgia
  - 205.452.01299 Boehringer Ingelheim Investigational Site, Gainesville, Georgia
  - 205.452.01288 Boehringer Ingelheim Investigational Site, Lawrenceville, Georgia
  - 205.452.01090 Boehringer Ingelheim Investigational Site, Snellville, Georgia
  - 205.452.01100 Boehringer Ingelheim Investigational Site, Honolulu, Hawaii
  - 205.452.01165 Boehringer Ingelheim Investigational Site, Boise, Idaho
  - 205.452.01059 Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - 205.452.01062 Boehringer Ingelheim Investigational Site, Eagle, Idaho
  - 205.452.01166 Boehringer Ingelheim Investigational Site, Hayden Lake, Idaho
  - 205.452.01275 Boehringer Ingelheim Investigational Site, Meridian, Idaho
  - 205.452.01330 Boehringer Ingelheim Investigational Site, Arlington Heights, Illinois
  - 205.452.01248 Boehringer Ingelheim Investigational Site, Belleville, Illinois
  - 205.452.01278 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 205.452.01371 Boehringer Ingelheim Investigational Site, Downer Grove, Illinois
  - 205.452.01235 Boehringer Ingelheim Investigational Site, Lombard, Illinois
  - 205.452.01180 Boehringer Ingelheim Investigational Site, O'Fallon, Illinois
  - 205.452.01268 Boehringer Ingelheim Investigational Site, Oak Park, Illinois
  - 205.452.01359 Boehringer Ingelheim Investigational Site, Quincy, Illinois
  - 205.452.01347 Boehringer Ingelheim Investigational Site, Brownsburg, Indiana
  - 205.452.01153 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 205.452.01301 Boehringer Ingelheim Investigational Site, Fishers, Indiana
  - 205.452.01141 Boehringer Ingelheim Investigational Site, Franklin, Indiana
  - 205.452.01137 Boehringer Ingelheim Investigational Site, Lafayette, Indiana
  - 205.452.01263 Boehringer Ingelheim Investigational Site, Muncie, Indiana
  - 205.452.01284 Boehringer Ingelheim Investigational Site, Council Bluffs, Iowa
  - 205.452.01021 Boehringer Ingelheim Investigational Site, Dubuque, Iowa
  - 205.452.01305 Boehringer Ingelheim Investigational Site, Lansing, Kansas
  - 205.452.01304 Boehringer Ingelheim Investigational Site, Olathe, Kansas
  - 205.452.01125 Boehringer Ingelheim Investigational Site, Overland Park, Kansas
  - 205.452.01068 Boehringer Ingelheim Investigational Site, Topeka, Kansas
  - 205.452.01063 Boehringer Ingelheim Investigational Site, Bowling Green, Kentucky
  - 205.452.01206 Boehringer Ingelheim Investigational Site, Fort Mitchell, Kentucky
  - 205.452.01289 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 205.452.01152 Boehringer Ingelheim Investigational Site, Paducah, Kentucky
  - 205.452.01015 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 205.452.01091 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 205.452.01329 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 205.452.01364 Boehringer Ingelheim Investigational Site, Auburn, Maine
  - 205.452.01169 Boehringer Ingelheim Investigational Site, Bangor, Maine
  - 205.452.01022 Boehringer Ingelheim Investigational Site, Biddeford, Maine
  - 205.452.01053 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 205.452.01190 Boehringer Ingelheim Investigational Site, Elkridge, Maryland
  - 205.452.01336 Boehringer Ingelheim Investigational Site, Hollywood, Maryland
  - 205.452.01238 Boehringer Ingelheim Investigational Site, Towson, Maryland
  - 205.452.01243 Boehringer Ingelheim Investigational Site, Towson, Maryland
  - 205.452.01366 Boehringer Ingelheim Investigational Site, Fall River, Massachusetts
  - 205.452.01269 Boehringer Ingelheim Investigational Site, Haverhill, Massachusetts
  - 205.452.01208 Boehringer Ingelheim Investigational Site, New Bedford, Massachusetts
  - 205.452.01170 Boehringer Ingelheim Investigational Site, Worcester, Massachusetts
  - 205.452.01270 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 205.452.01349 Boehringer Ingelheim Investigational Site, Benzonia, Michigan
  - 205.452.01365 Boehringer Ingelheim Investigational Site, Chelsea, Michigan
  - 205.452.01149 Boehringer Ingelheim Investigational Site, Chesterfield, Michigan
  - 205.452.01146 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 205.452.01139 Boehringer Ingelheim Investigational Site, Interlochen, Michigan
  - 205.452.01080 Boehringer Ingelheim Investigational Site, Kalamazoo, Michigan
  - 205.452.01310 Boehringer Ingelheim Investigational Site, Stevensville, Michigan
  - 205.452.01122 Boehringer Ingelheim Investigational Site, Traverse City, Michigan
  - 205.452.01081 Boehringer Ingelheim Investigational Site, Troy, Michigan
  - 205.452.01221 Boehringer Ingelheim Investigational Site, Troy, Michigan
  - 205.452.01205 Boehringer Ingelheim Investigational Site, Chaska, Minnesota
  - 205.452.01211 Boehringer Ingelheim Investigational Site, Edina, Minnesota
  - 205.452.01104 Boehringer Ingelheim Investigational Site, Fridley, Minnesota
  - 205.452.01113 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 205.452.01042 Boehringer Ingelheim Investigational Site, Rochester, Minnesota
  - 205.452.01019 Boehringer Ingelheim Investigational Site, Olive Branch, Mississippi
  - 205.452.01014 Boehringer Ingelheim Investigational Site, Chesterfield, Missouri
  - 205.452.01129 Boehringer Ingelheim Investigational Site, Saint Charles, Missouri
  - 205.452.01110 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 205.452.01179 Boehringer Ingelheim Investigational Site, West Plains, Missouri
  - 205.452.01226 Boehringer Ingelheim Investigational Site, Billings, Montana
  - 205.452.01076 Boehringer Ingelheim Investigational Site, Butte, Montana
  - 205.452.01196 Boehringer Ingelheim Investigational Site, Missoula, Montana
  - 205.452.01150 Boehringer Ingelheim Investigational Site, Bellevue, Nebraska
  - 205.452.01187 Boehringer Ingelheim Investigational Site, Fremont, Nebraska
  - 205.452.01155 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 205.452.01073 Boehringer Ingelheim Investigational Site, Henderson, Nevada
  - 205.452.01031 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 205.452.01261 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 205.452.01026 Boehringer Ingelheim Investigational Site, Lebanon, New Hampshire
  - 205.452.01369 Boehringer Ingelheim Investigational Site, Newington, New Hampshire
  - 205.452.01296 Boehringer Ingelheim Investigational Site, Ocean City, New Jersey
  - 205.452.01046 Boehringer Ingelheim Investigational Site, Toms River, New Jersey
  - 205.452.01061 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 205.452.01167 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 205.452.01159 Boehringer Ingelheim Investigational Site, Bayside, New York
  - 205.452.01163 Boehringer Ingelheim Investigational Site, Bronxville, New York
  - 205.452.01194 Boehringer Ingelheim Investigational Site, Cooperstown, New York
  - 205.452.01131 Boehringer Ingelheim Investigational Site, Elmira, New York
  - 205.452.01142 Boehringer Ingelheim Investigational Site, Endwell, New York
  - 205.452.01192 Boehringer Ingelheim Investigational Site, Glens Falls, New York
  - 205.452.01279 Boehringer Ingelheim Investigational Site, Great Neck, New York
  - 205.452.01328 Boehringer Ingelheim Investigational Site, Honeoye Falls, New York
  - 205.452.01118 Boehringer Ingelheim Investigational Site, New Windsor, New York
  - 205.452.01127 Boehringer Ingelheim Investigational Site, New York, New York
  - 205.452.01058 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 205.452.01085 Boehringer Ingelheim Investigational Site, Syracuse, New York
  - 205.452.01293 Boehringer Ingelheim Investigational Site, Syracuse, New York
  - 205.452.01151 Boehringer Ingelheim Investigational Site, Vestal, New York
  - 205.452.01188 Boehringer Ingelheim Investigational Site, Westfield, New York
  - 205.452.01271 Boehringer Ingelheim Investigational Site, Asheville, North Carolina
  - 205.452.01101 Boehringer Ingelheim Investigational Site, Burlington, North Carolina
  - 205.452.01264 Boehringer Ingelheim Investigational Site, Calabash, North Carolina
  - 205.452.01168 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 205.452.01108 Boehringer Ingelheim Investigational Site, Elizabeth City, North Carolina
  - 205.452.01033 Boehringer Ingelheim Investigational Site, Greensboro, North Carolina
  - 205.452.01172 Boehringer Ingelheim Investigational Site, Greensboro, North Carolina
  - 205.452.01098 Boehringer Ingelheim Investigational Site, Hickory, North Carolina
  - 205.452.01115 Boehringer Ingelheim Investigational Site, Hickory, North Carolina
  - 205.452.01128 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 205.452.01352 Boehringer Ingelheim Investigational Site, Rocky Mount, North Carolina
  - 205.452.01348 Boehringer Ingelheim Investigational Site, Salisbury, North Carolina
  - 205.452.01032 Boehringer Ingelheim Investigational Site, Statesville, North Carolina
  - 205.452.01276 Boehringer Ingelheim Investigational Site, Tabor City, North Carolina
  - 205.452.01157 Boehringer Ingelheim Investigational Site, Wilmington, North Carolina
  - 205.452.01363 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 205.452.01193 Boehringer Ingelheim Investigational Site, Canal Fulton, Ohio
  - 205.452.01374 Boehringer Ingelheim Investigational Site, Centerville, Ohio
  - 205.452.01006 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 205.452.01373 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 205.452.01314 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 205.452.01210 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 205.452.01232 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 205.452.01309 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 205.452.01140 Boehringer Ingelheim Investigational Site, Delaware, Ohio
  - 205.452.01084 Boehringer Ingelheim Investigational Site, Sylvania, Ohio
  - 205.452.01287 Boehringer Ingelheim Investigational Site, Toledo, Ohio
  - 205.452.01010 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 205.452.01094 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 205.452.01029 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 205.452.01043 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 205.452.01266 Boehringer Ingelheim Investigational Site, Ashland, Oregon
  - 205.452.01083 Boehringer Ingelheim Investigational Site, Bend, Oregon
  - 205.452.01189 Boehringer Ingelheim Investigational Site, Corvallis, Oregon
  - 205.452.01341 Boehringer Ingelheim Investigational Site, Springfield, Oregon
  - 205.452.01002 Boehringer Ingelheim Investigational Site, Altoona, Pennsylvania
  - 205.452.01354 Boehringer Ingelheim Investigational Site, Beaver, Pennsylvania
  - 205.452.01143 Boehringer Ingelheim Investigational Site, Carnegie, Pennsylvania
  - 205.452.01320 Boehringer Ingelheim Investigational Site, Downingtown, Pennsylvania
  - 205.452.01323 Boehringer Ingelheim Investigational Site, Erie, Pennsylvania
  - 205.452.01257 Boehringer Ingelheim Investigational Site, Jefferson Hills, Pennsylvania
  - 205.452.01332 Boehringer Ingelheim Investigational Site, Langhorne, Pennsylvania
  - 205.452.01075 Boehringer Ingelheim Investigational Site, Norristown, Pennsylvania
  - 205.452.01087 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 205.452.01144 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 205.452.01003 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 205.452.01361 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 205.452.01036 Boehringer Ingelheim Investigational Site, Pleasant Hills, Pennsylvania
  - 205.452.01106 Boehringer Ingelheim Investigational Site, Uniontown, Pennsylvania
  - 205.452.01156 Boehringer Ingelheim Investigational Site, Uniontown, Pennsylvania
  - 205.452.01204 Boehringer Ingelheim Investigational Site, Warminster, Pennsylvania
  - 205.452.01338 Boehringer Ingelheim Investigational Site, Wyomissing, Pennsylvania
  - 205.452.01267 Boehringer Ingelheim Investigational Site, Cranston, Rhode Island
  - 205.452.01214 Boehringer Ingelheim Investigational Site, Johnston, Rhode Island
  - 205.452.01340 Boehringer Ingelheim Investigational Site, Anderson, South Carolina
  - 205.452.01066 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 205.452.01217 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 205.452.01303 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 205.452.01259 Boehringer Ingelheim Investigational Site, Florence, South Carolina
  - 205.452.01013 Boehringer Ingelheim Investigational Site, Gaffney, South Carolina
  - 205.452.01077 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 205.452.01093 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 205.452.01295 Boehringer Ingelheim Investigational Site, Hodges, South Carolina
  - 205.452.01335 Boehringer Ingelheim Investigational Site, Myrtle Beach, South Carolina
  - 205.452.01056 Boehringer Ingelheim Investigational Site, Rock Hill, South Carolina
  - 205.452.01294 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 205.452.01004 Boehringer Ingelheim Investigational Site, Rapid City, South Dakota
  - 205.452.01126 Boehringer Ingelheim Investigational Site, Brentwood, Tennessee
  - 205.452.01220 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 205.452.01324 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 205.452.01342 Boehringer Ingelheim Investigational Site, Kingsport, Tennessee
  - 205.452.01096 Boehringer Ingelheim Investigational Site, Arlington, Texas
  - 205.452.01050 Boehringer Ingelheim Investigational Site, Corsicana, Texas
  - 205.452.01233 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 205.452.01334 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 205.452.01057 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 205.452.01181 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 205.452.01272 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 205.452.01082 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 205.452.01105 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 205.452.01178 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 205.452.01212 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 205.452.01274 Boehringer Ingelheim Investigational Site, Longview, Texas
  - 205.452.01116 Boehringer Ingelheim Investigational Site, McKinney, Texas
  - 205.452.01262 Boehringer Ingelheim Investigational Site, Richardson, Texas
  - 205.452.01055 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 205.452.01182 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 205.452.01186 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 205.452.01353 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 205.452.01215 Boehringer Ingelheim Investigational Site, Sugar Land, Texas
  - 205.452.01223 Boehringer Ingelheim Investigational Site, Midvale, Utah
  - 205.452.01001 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 205.452.01079 Boehringer Ingelheim Investigational Site, Abingdon, Virginia
  - 205.452.01234 Boehringer Ingelheim Investigational Site, Alexandria, Virginia
  - 205.452.01065 Boehringer Ingelheim Investigational Site, Danville, Virginia
  - 205.452.01285 Boehringer Ingelheim Investigational Site, Danville, Virginia
  - 205.452.01045 Boehringer Ingelheim Investigational Site, Ettrick, Virginia
  - 205.452.01030 Boehringer Ingelheim Investigational Site, Lynchburg, Virginia
  - 205.452.01016 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 205.452.01039 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 205.452.01044 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 205.452.01300 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 205.452.01099 Boehringer Ingelheim Investigational Site, Selah, Washington
  - 205.452.01008 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 205.452.01069 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 205.452.01145 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 205.452.01185 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 205.452.01007 Boehringer Ingelheim Investigational Site, Wenatchee, Washington
  - 205.452.01201 Boehringer Ingelheim Investigational Site, Oregon, Wisconsin
  - 205.452.01344 Boehringer Ingelheim Investigational Site, West Allis, Wisconsin
- Argentina (16):
  - 205.452.54003 Boehringer Ingelheim Investigational Site, Capital Federal
  - 205.452.54011 Boehringer Ingelheim Investigational Site, Capital Federal
  - 205.452.54013 Boehringer Ingelheim Investigational Site, Capital Federal
  - 205.452.54027 Boehringer Ingelheim Investigational Site, Capital Federal
  - 205.452.54029 Boehringer Ingelheim Investigational Site, Capital Federal
  - 205.452.54031 Boehringer Ingelheim Investigational Site, Capital Federal
  - 205.452.54007 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 205.452.54015 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 205.452.54001 Boehringer Ingelheim Investigational Site, Mendoza
  - 205.452.54019 Boehringer Ingelheim Investigational Site, Monte Grande
  - 205.452.54005 Boehringer Ingelheim Investigational Site, Quilmes
  - 205.452.54009 Boehringer Ingelheim Investigational Site, Rosario
  - 205.452.54021 Boehringer Ingelheim Investigational Site, Rosario
  - 205.452.54025 Boehringer Ingelheim Investigational Site, San Juan Bautista
  - 205.452.54017 Boehringer Ingelheim Investigational Site, San Miguel de Tucumán
  - 205.452.54023 Boehringer Ingelheim Investigational Site, San Miguel de Tucumán
- Australia (6):
  - 205.452.61006 Boehringer Ingelheim Investigational Site, Adelaide, South Australia
  - 205.452.61002 Boehringer Ingelheim Investigational Site, Woodville, South Australia
  - 205.452.61004 Boehringer Ingelheim Investigational Site, Box Hill, Victoria
  - 205.452.61003 Boehringer Ingelheim Investigational Site, Footscray, Victoria
  - 205.452.61001 Boehringer Ingelheim Investigational Site, Frankston, Victoria
  - 205.452.61005 Boehringer Ingelheim Investigational Site, Nedlands, Western Australia
- Austria (3):
  - 205.452.43002 Boehringer Ingelheim Investigational Site, Feldbach
  - 205.452.43003 Boehringer Ingelheim Investigational Site, Hallein
  - 205.452.43005 Boehringer Ingelheim Investigational Site, Thalheim bei Wels
- Belgium (9):
  - 205.452.32009 Boehringer Ingelheim Investigational Site, Godinne
  - 205.452.32007 Boehringer Ingelheim Investigational Site, Gozée
  - 205.452.32002 Boehringer Ingelheim Investigational Site, Halen
  - 205.452.32001 Boehringer Ingelheim Investigational Site, Leuven
  - 205.452.32006 Boehringer Ingelheim Investigational Site, Linkebeek
  - 205.452.32005 Boehringer Ingelheim Investigational Site, Merksem
  - 205.452.32008 Boehringer Ingelheim Investigational Site, Natoye
  - 205.452.32003 Boehringer Ingelheim Investigational Site, Tessenderlo
  - 205.452.32004 Boehringer Ingelheim Investigational Site, Zichem
- Brazil (11):
  - 205.452.55005 Boehringer Ingelheim Investigational Site, Florianópolis
  - 205.452.55010 Boehringer Ingelheim Investigational Site, Passo Fundo - RS
  - 205.452.55001 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 205.452.55002 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 205.452.55003 Boehringer Ingelheim Investigational Site, Recife
  - 205.452.55004 Boehringer Ingelheim Investigational Site, Rio de Janeiro
  - 205.452.55011 Boehringer Ingelheim Investigational Site, Rio de Janeiro
  - 205.452.55008 Boehringer Ingelheim Investigational Site, Sao Pablo
  - 205.452.55006 Boehringer Ingelheim Investigational Site, São Paulo
  - 205.452.55007 Boehringer Ingelheim Investigational Site, São Paulo
  - 205.452.55009 Boehringer Ingelheim Investigational Site, São Paulo
- Bulgaria (12):
  - 205.452.35909 Boehringer Ingelheim Investigational Site, Plovdiv
  - 205.452.35910 Boehringer Ingelheim Investigational Site, Plovdiv
  - 205.452.35901 Boehringer Ingelheim Investigational Site, Sofia
  - 205.452.35902 Boehringer Ingelheim Investigational Site, Sofia
  - 205.452.35903 Boehringer Ingelheim Investigational Site, Sofia
  - 205.452.35904 Boehringer Ingelheim Investigational Site, Sofia
  - 205.452.35905 Boehringer Ingelheim Investigational Site, Sofia
  - 205.452.35908 Boehringer Ingelheim Investigational Site, Sofia
  - 205.452.35914 Boehringer Ingelheim Investigational Site, Sofia
  - 205.452.35915 Boehringer Ingelheim Investigational Site, Sofia
  - 205.452.35912 Boehringer Ingelheim Investigational Site, Stara Zagora
  - 205.452.35906 Boehringer Ingelheim Investigational Site, Veliko Tarnovo
- Canada (50):
  - 205.452.11015 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 205.452.11032 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 205.452.11028 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 205.452.11037 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 205.452.11045 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 205.452.11047 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 205.452.11002 Boehringer Ingelheim Investigational Site, Spruce Grove, Alberta
  - 205.452.11048 Boehringer Ingelheim Investigational Site, Kelowna, British Columbia
  - 205.452.11051 Boehringer Ingelheim Investigational Site, Maple Ridge, British Columbia
  - 205.452.11014 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 205.452.11016 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 205.452.11025 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 205.452.11033 Boehringer Ingelheim Investigational Site, Moncton, New Brunswick
  - 205.452.11010 Boehringer Ingelheim Investigational Site, Saint John, New Brunswick
  - 205.452.11044 Boehringer Ingelheim Investigational Site, Grand Falls-Windsor, Newfoundland and Labrador
  - 205.452.11053 Boehringer Ingelheim Investigational Site, Mount Pearl, Newfoundland and Labrador
  - 205.452.11017 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 205.452.11021 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 205.452.11030 Boehringer Ingelheim Investigational Site, Burlington, Ontario
  - 205.452.11042 Boehringer Ingelheim Investigational Site, Corunna, Ontario
  - 205.452.11049 Boehringer Ingelheim Investigational Site, Courtice, Ontario
  - 205.452.11004 Boehringer Ingelheim Investigational Site, Downsview, Ontario
  - 205.452.11009 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 205.452.11029 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 205.452.11050 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 205.452.11040 Boehringer Ingelheim Investigational Site, Kingston, Ontario
  - 205.452.11035 Boehringer Ingelheim Investigational Site, London, Ontario
  - 205.452.11001 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 205.452.11054 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 205.452.11022 Boehringer Ingelheim Investigational Site, Newmarket, Ontario
  - 205.452.11024 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 205.452.11027 Boehringer Ingelheim Investigational Site, Richmond Hill, Ontario
  - 205.452.11041 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 205.452.11019 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 205.452.11034 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 205.452.11052 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 205.452.11012 Boehringer Ingelheim Investigational Site, Windsor, Ontario
  - 205.452.11007 Boehringer Ingelheim Investigational Site, Greenfield Park, Quebec
  - 205.452.11005 Boehringer Ingelheim Investigational Site, La Malbaie, Quebec
  - 205.452.11006 Boehringer Ingelheim Investigational Site, Longueuil, Quebec
  - 205.452.11043 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 205.452.11013 Boehringer Ingelheim Investigational Site, Point Claire, Quebec
  - 205.452.11031 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 205.452.11020 Boehringer Ingelheim Investigational Site, Saint-Lambert, Quebec
  - 205.452.11018 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
  - 205.452.11026 Boehringer Ingelheim Investigational Site, Trois-Rivières, Quebec
  - 205.452.11003 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
  - 205.452.11011 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
  - 205.452.11036 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
  - 205.452.11039 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- China (36):
  - 205.452.86009 Boehringer Ingelheim Investigational Site, Beijing
  - 205.452.86010 Boehringer Ingelheim Investigational Site, Beijing
  - 205.452.86011 Boehringer Ingelheim Investigational Site, Beijing
  - 205.452.86012 Boehringer Ingelheim Investigational Site, Beijing
  - 205.452.86038 Boehringer Ingelheim Investigational Site, Beijing
  - 205.452.86026 Boehringer Ingelheim Investigational Site, Changchun
  - 205.452.86024 Boehringer Ingelheim Investigational Site, Changsha
  - 205.452.86025 Boehringer Ingelheim Investigational Site, Changsha
  - 205.452.86021 Boehringer Ingelheim Investigational Site, Chengdu
  - 205.452.86032 Boehringer Ingelheim Investigational Site, Chengdu
  - 205.452.86034 Boehringer Ingelheim Investigational Site, Chongqing
  - 205.452.86035 Boehringer Ingelheim Investigational Site, Chongqing
  - 205.452.86036 Boehringer Ingelheim Investigational Site, Chongqing
  - 205.452.86020 Boehringer Ingelheim Investigational Site, Foshan
  - 205.452.86001 Boehringer Ingelheim Investigational Site, Guangzhou
  - 205.452.86004 Boehringer Ingelheim Investigational Site, Guangzhou
  - 205.452.86005 Boehringer Ingelheim Investigational Site, Guangzhou
  - 205.452.86019 Boehringer Ingelheim Investigational Site, Guangzhou
  - 205.452.86028 Boehringer Ingelheim Investigational Site, Guangzhou
  - 205.452.86030 Boehringer Ingelheim Investigational Site, Haikou
  - 205.452.86007 Boehringer Ingelheim Investigational Site, Hangzhou
  - 205.452.86008 Boehringer Ingelheim Investigational Site, Hangzhou
  - 205.452.86037 Boehringer Ingelheim Investigational Site, Nanchang
  - 205.452.86022 Boehringer Ingelheim Investigational Site, Nanjing
  - 205.452.86029 Boehringer Ingelheim Investigational Site, Nanning
  - 205.452.86027 Boehringer Ingelheim Investigational Site, Qingdao
  - 205.452.86002 Boehringer Ingelheim Investigational Site, Shanghai
  - 205.452.86003 Boehringer Ingelheim Investigational Site, Shanghai
  - 205.452.86018 Boehringer Ingelheim Investigational Site, Shanghai
  - 205.452.86014 Boehringer Ingelheim Investigational Site, Shenyang
  - 205.452.86015 Boehringer Ingelheim Investigational Site, Shenyang
  - 205.452.86006 Boehringer Ingelheim Investigational Site, Suzhou
  - 205.452.86033 Boehringer Ingelheim Investigational Site, Tianjin
  - 205.452.86031 Boehringer Ingelheim Investigational Site, Wuhan
  - 205.452.86016 Boehringer Ingelheim Investigational Site, Xi'an
  - 205.452.86017 Boehringer Ingelheim Investigational Site, Xi'an
- Colombia (5):
  - 205.452.57002 Boehringer Ingelheim Investigational Site, Bogotá
  - 205.452.57004 Boehringer Ingelheim Investigational Site, Bogotá
  - 205.452.57005 Boehringer Ingelheim Investigational Site, Bogotá
  - 205.452.57006 Boehringer Ingelheim Investigational Site, Bogotá
  - 205.452.57001 Boehringer Ingelheim Investigational Site, Medellín
- Croatia (12):
  - 205.452.38512 Boehringer Ingelheim Investigational Site, Čakovec
  - 205.452.38508 Boehringer Ingelheim Investigational Site, Dubrovnik
  - 205.452.38510 Boehringer Ingelheim Investigational Site, Osijek
  - 205.452.38501 Boehringer Ingelheim Investigational Site, Rijeka
  - 205.452.38506 Boehringer Ingelheim Investigational Site, Sisak
  - 205.452.38502 Boehringer Ingelheim Investigational Site, Split
  - 205.452.38503 Boehringer Ingelheim Investigational Site, Split
  - 205.452.38504 Boehringer Ingelheim Investigational Site, Zagreb
  - 205.452.38505 Boehringer Ingelheim Investigational Site, Zagreb
  - 205.452.38507 Boehringer Ingelheim Investigational Site, Zagreb
  - 205.452.38509 Boehringer Ingelheim Investigational Site, Zagreb
  - 205.452.38511 Boehringer Ingelheim Investigational Site, Zagreb
- Denmark (15):
  - 205.452.45002 Boehringer Ingelheim Investigational Site, Aalborg
  - 205.452.45003 Boehringer Ingelheim Investigational Site, Aarhus C
  - 205.452.45006 Boehringer Ingelheim Investigational Site, Birkerød
  - 205.452.45013 Boehringer Ingelheim Investigational Site, Kolding
  - 205.452.45001 Boehringer Ingelheim Investigational Site, København NV
  - 205.452.45005 Boehringer Ingelheim Investigational Site, København S
  - 205.452.45012 Boehringer Ingelheim Investigational Site, Odense C
  - 205.452.45016 Boehringer Ingelheim Investigational Site, Roskilde
  - 205.452.45009 Boehringer Ingelheim Investigational Site, Rødovre Municipality
  - 205.452.45010 Boehringer Ingelheim Investigational Site, Rødovre Municipality
  - 205.452.45004 Boehringer Ingelheim Investigational Site, Silkeborg
  - 205.452.45014 Boehringer Ingelheim Investigational Site, Skive
  - 205.452.45011 Boehringer Ingelheim Investigational Site, Sønderborg
  - 205.452.45015 Boehringer Ingelheim Investigational Site, Viby J
  - 205.452.45007 Boehringer Ingelheim Investigational Site, Værløse
- Finland (7):
  - 205.452.35806 Boehringer Ingelheim Investigational Site, Ekenäs
  - 205.452.35801 Boehringer Ingelheim Investigational Site, Helsinki
  - 205.452.35804 Boehringer Ingelheim Investigational Site, Lahti
  - 205.452.35808 Boehringer Ingelheim Investigational Site, Pori
  - 205.452.35805 Boehringer Ingelheim Investigational Site, Porvoo
  - 205.452.35802 Boehringer Ingelheim Investigational Site, Tampere
  - 205.452.35803 Boehringer Ingelheim Investigational Site, Turku
- France (94):
  - 205.452.33087 Boehringer Ingelheim Investigational Site, Albens
  - 205.452.33028 Boehringer Ingelheim Investigational Site, Angers
  - 205.452.33055 Boehringer Ingelheim Investigational Site, Angers
  - 205.452.33142 Boehringer Ingelheim Investigational Site, Angers
  - 205.452.33159 Boehringer Ingelheim Investigational Site, Angers
  - 205.452.33030 Boehringer Ingelheim Investigational Site, Anzin
  - 205.452.33158 Boehringer Ingelheim Investigational Site, Arras
  - 205.452.33084 Boehringer Ingelheim Investigational Site, Avrillé
  - 205.452.33029 Boehringer Ingelheim Investigational Site, Bersée
  - 205.452.33128 Boehringer Ingelheim Investigational Site, Bécon-les-Granits
  - 205.452.33018 Boehringer Ingelheim Investigational Site, Béziers
  - 205.452.33053 Boehringer Ingelheim Investigational Site, Bischheim
  - 205.452.33024 Boehringer Ingelheim Investigational Site, Blois
  - 205.452.33043 Boehringer Ingelheim Investigational Site, Bort-les-Orgues
  - 205.452.33091 Boehringer Ingelheim Investigational Site, Bourg Des Cptes
  - 205.452.33123 Boehringer Ingelheim Investigational Site, Briollay
  - 205.452.33063 Boehringer Ingelheim Investigational Site, Broglie
  - 205.452.33074 Boehringer Ingelheim Investigational Site, Bruay-la-Buissière
  - 205.452.33010 Boehringer Ingelheim Investigational Site, Cannes
  - 205.452.33118 Boehringer Ingelheim Investigational Site, Cannes
  - 205.452.33009 Boehringer Ingelheim Investigational Site, Chamalières
  - 205.452.33073 Boehringer Ingelheim Investigational Site, Chambéry
  - 205.452.33059 Boehringer Ingelheim Investigational Site, Château-Renault
  - 205.452.33089 Boehringer Ingelheim Investigational Site, Colombey-les-Belles
  - 205.452.33099 Boehringer Ingelheim Investigational Site, Cournonterral
  - 205.452.33127 Boehringer Ingelheim Investigational Site, Cournonterral
  - 205.452.33162 Boehringer Ingelheim Investigational Site, Croix
  - 205.452.33105 Boehringer Ingelheim Investigational Site, Dinard
  - 205.452.33110 Boehringer Ingelheim Investigational Site, Donges
  - 205.452.33094 Boehringer Ingelheim Investigational Site, Gambsheim
  - 205.452.33046 Boehringer Ingelheim Investigational Site, Grenoble
  - 205.452.33096 Boehringer Ingelheim Investigational Site, Hautmont
  - 205.452.33090 Boehringer Ingelheim Investigational Site, Hinx
  - 205.452.33145 Boehringer Ingelheim Investigational Site, Jarny
  - 205.452.33154 Boehringer Ingelheim Investigational Site, La Bouëxière
  - 205.452.33065 Boehringer Ingelheim Investigational Site, La Chapelle-sur-Erdre
  - 205.452.33102 Boehringer Ingelheim Investigational Site, La Montagne
  - 205.452.33100 Boehringer Ingelheim Investigational Site, La Riche
  - 205.452.33058 Boehringer Ingelheim Investigational Site, Lambersart
  - 205.452.33098 Boehringer Ingelheim Investigational Site, Lambersart
  - 205.452.33103 Boehringer Ingelheim Investigational Site, Levallois-Perret
  - 205.452.33164 Boehringer Ingelheim Investigational Site, Louvigné-de-Bais
  - 205.452.33111 Boehringer Ingelheim Investigational Site, Luynes
  - 205.452.33136 Boehringer Ingelheim Investigational Site, Marcq-en-Barœul
  - 205.452.33115 Boehringer Ingelheim Investigational Site, Mondelange
  - 205.452.33088 Boehringer Ingelheim Investigational Site, Mont-de-Marsan
  - 205.452.33138 Boehringer Ingelheim Investigational Site, Mont-de-Marsan
  - 205.452.33005 Boehringer Ingelheim Investigational Site, Montigny-lès-Metz
  - 205.452.33163 Boehringer Ingelheim Investigational Site, Mundolsheim
  - 205.452.33109 Boehringer Ingelheim Investigational Site, Mûrs-Erigné
  - 205.452.33031 Boehringer Ingelheim Investigational Site, Nantes
  - 205.452.33003 Boehringer Ingelheim Investigational Site, Nice
  - 205.452.33108 Boehringer Ingelheim Investigational Site, Oignies
  - 205.452.33014 Boehringer Ingelheim Investigational Site, Ollioules
  - 205.452.33157 Boehringer Ingelheim Investigational Site, Orthez
  - 205.452.33112 Boehringer Ingelheim Investigational Site, Parçay-les-Pins
  - 205.452.33001 Boehringer Ingelheim Investigational Site, Paris
  - 205.452.33051 Boehringer Ingelheim Investigational Site, Paris
  - 205.452.33082 Boehringer Ingelheim Investigational Site, Paris
  - 205.452.33165 Boehringer Ingelheim Investigational Site, Paris
  - 205.452.33130 Boehringer Ingelheim Investigational Site, Pont-à-Mousson
  - 205.452.33122 Boehringer Ingelheim Investigational Site, Quarouble
  - 205.452.33006 Boehringer Ingelheim Investigational Site, Reims
  - 205.452.33153 Boehringer Ingelheim Investigational Site, Rosiers-d'Égletons
  - 205.452.33161 Boehringer Ingelheim Investigational Site, Rugles
  - 205.452.33126 Boehringer Ingelheim Investigational Site, Saint-Alban-Leysse
  - 205.452.33140 Boehringer Ingelheim Investigational Site, Saint-Aulaire
  - 205.452.33052 Boehringer Ingelheim Investigational Site, Saint-Avertin
  - 205.452.33160 Boehringer Ingelheim Investigational Site, Saint-Jouan-des-Guérets
  - 205.452.33011 Boehringer Ingelheim Investigational Site, Saint-Léger-des-Bois
  - 205.452.33079 Boehringer Ingelheim Investigational Site, Saint-Sébastien-sur-Loire
  - 205.452.33002 Boehringer Ingelheim Investigational Site, Saintes
  - 205.452.33148 Boehringer Ingelheim Investigational Site, Salies-de-Béarn
  - 205.452.33026 Boehringer Ingelheim Investigational Site, Savonnières
  - 205.452.33067 Boehringer Ingelheim Investigational Site, Segré
  - 205.452.33040 Boehringer Ingelheim Investigational Site, Serres Casset
  - 205.452.33012 Boehringer Ingelheim Investigational Site, Six Four Les Plages
  - 205.452.33007 Boehringer Ingelheim Investigational Site, Strasbourg
  - 205.452.33033 Boehringer Ingelheim Investigational Site, Strasbourg
  - 205.452.33097 Boehringer Ingelheim Investigational Site, Strasbourg
  - 205.452.33101 Boehringer Ingelheim Investigational Site, Strasbourg
  - 205.452.33107 Boehringer Ingelheim Investigational Site, Thouars
  - 205.452.33116 Boehringer Ingelheim Investigational Site, Tinténiac
  - 205.452.33013 Boehringer Ingelheim Investigational Site, Toulon
  - 205.452.33054 Boehringer Ingelheim Investigational Site, Tours
  - 205.452.33064 Boehringer Ingelheim Investigational Site, Tours
  - 205.452.33092 Boehringer Ingelheim Investigational Site, Tours
  - 205.452.33124 Boehringer Ingelheim Investigational Site, Tours
  - 205.452.33066 Boehringer Ingelheim Investigational Site, Vendôme
  - 205.452.33137 Boehringer Ingelheim Investigational Site, Vernoil-le-Fourrier
  - 205.452.33032 Boehringer Ingelheim Investigational Site, Vieux-Condé
  - 205.452.33151 Boehringer Ingelheim Investigational Site, Vihiers
  - 205.452.33077 Boehringer Ingelheim Investigational Site, Villey-Saint-Étienne
  - 205.452.33135 Boehringer Ingelheim Investigational Site, Wattrelos
- Georgia (7):
  - 205.452.99501 Boehringer Ingelheim Investigational Site, Tbilisi
  - 205.452.99502 Boehringer Ingelheim Investigational Site, Tbilisi
  - 205.452.99503 Boehringer Ingelheim Investigational Site, Tbilisi
  - 205.452.99504 Boehringer Ingelheim Investigational Site, Tbilisi
  - 205.452.99505 Boehringer Ingelheim Investigational Site, Tbilisi
  - 205.452.99506 Boehringer Ingelheim Investigational Site, Tbilisi
  - 205.452.99507 Boehringer Ingelheim Investigational Site, Tbilisi
- Germany (115):
  - 205.452.49096 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 205.452.49130 Boehringer Ingelheim Investigational Site, Augsburg
  - 205.452.49161 Boehringer Ingelheim Investigational Site, Augsburg
  - 205.452.49001 Boehringer Ingelheim Investigational Site, Backnang
  - 205.452.49173 Boehringer Ingelheim Investigational Site, Bad Kissingen
  - 205.452.49134 Boehringer Ingelheim Investigational Site, Bad Lippspringe
  - 205.452.49082 Boehringer Ingelheim Investigational Site, Bad Neustadt an der Saale
  - 205.452.49058 Boehringer Ingelheim Investigational Site, Bad Wörishofen
  - 205.452.49145 Boehringer Ingelheim Investigational Site, Bamberg
  - 205.452.49072 Boehringer Ingelheim Investigational Site, Bensheim
  - 205.452.49048 Boehringer Ingelheim Investigational Site, Bergisch Gladbach
  - 205.452.49006 Boehringer Ingelheim Investigational Site, Berlin
  - 205.452.49016 Boehringer Ingelheim Investigational Site, Berlin
  - 205.452.49028 Boehringer Ingelheim Investigational Site, Berlin
  - 205.452.49031 Boehringer Ingelheim Investigational Site, Berlin
  - 205.452.49054 Boehringer Ingelheim Investigational Site, Berlin
  - 205.452.49064 Boehringer Ingelheim Investigational Site, Berlin
  - 205.452.49066 Boehringer Ingelheim Investigational Site, Berlin
  - 205.452.49068 Boehringer Ingelheim Investigational Site, Berlin
  - 205.452.49102 Boehringer Ingelheim Investigational Site, Berlin
  - 205.452.49135 Boehringer Ingelheim Investigational Site, Berlin
  - 205.452.49138 Boehringer Ingelheim Investigational Site, Berlin
  - 205.452.49157 Boehringer Ingelheim Investigational Site, Berlin
  - 205.452.49167 Boehringer Ingelheim Investigational Site, Berlin
  - 205.452.49175 Boehringer Ingelheim Investigational Site, Berlin
  - 205.452.49180 Boehringer Ingelheim Investigational Site, Berlin
  - 205.452.49037 Boehringer Ingelheim Investigational Site, Bonn
  - 205.452.49118 Boehringer Ingelheim Investigational Site, Bonn
  - 205.452.49083 Boehringer Ingelheim Investigational Site, Brake
  - 205.452.49040 Boehringer Ingelheim Investigational Site, Bruchsal
  - 205.452.49089 Boehringer Ingelheim Investigational Site, Celle
  - 205.452.49146 Boehringer Ingelheim Investigational Site, Cologne
  - 205.452.49143 Boehringer Ingelheim Investigational Site, Cottbus
  - 205.452.49119 Boehringer Ingelheim Investigational Site, Deggendorf
  - 205.452.49151 Boehringer Ingelheim Investigational Site, Dillingen
  - 205.452.49117 Boehringer Ingelheim Investigational Site, Donaueschingen
  - 205.452.49015 Boehringer Ingelheim Investigational Site, Dortmund
  - 205.452.49008 Boehringer Ingelheim Investigational Site, Düren
  - 205.452.49098 Boehringer Ingelheim Investigational Site, Emden
  - 205.452.49003 Boehringer Ingelheim Investigational Site, Engelskirchen
  - 205.452.49024 Boehringer Ingelheim Investigational Site, Ense
  - 205.452.49168 Boehringer Ingelheim Investigational Site, Essen
  - 205.452.49104 Boehringer Ingelheim Investigational Site, Forchheim
  - 205.452.49133 Boehringer Ingelheim Investigational Site, Föhren
  - 205.452.49070 Boehringer Ingelheim Investigational Site, Frankfurt
  - 205.452.49147 Boehringer Ingelheim Investigational Site, Frankfurt
  - 205.452.49137 Boehringer Ingelheim Investigational Site, Fulda
  - 205.452.49107 Boehringer Ingelheim Investigational Site, Gelnhausen
  - 205.452.49032 Boehringer Ingelheim Investigational Site, Gütersloh
  - 205.452.49026 Boehringer Ingelheim Investigational Site, Hagen
  - 205.452.49041 Boehringer Ingelheim Investigational Site, Hagen
  - 205.452.49044 Boehringer Ingelheim Investigational Site, Hamburg
  - 205.452.49061 Boehringer Ingelheim Investigational Site, Hamburg
  - 205.452.49080 Boehringer Ingelheim Investigational Site, Hamburg
  - 205.452.49038 Boehringer Ingelheim Investigational Site, Hanover
  - 205.452.49052 Boehringer Ingelheim Investigational Site, Hanover
  - 205.452.49094 Boehringer Ingelheim Investigational Site, Hanover
  - 205.452.49181 Boehringer Ingelheim Investigational Site, Heidelberg
  - 205.452.49116 Boehringer Ingelheim Investigational Site, Heilbronn
  - 205.452.49022 Boehringer Ingelheim Investigational Site, Hemmingen
  - 205.452.49007 Boehringer Ingelheim Investigational Site, Höchstädt
  - 205.452.49136 Boehringer Ingelheim Investigational Site, Ingelheim
  - 205.452.49159 Boehringer Ingelheim Investigational Site, Karlsruhe
  - 205.452.49027 Boehringer Ingelheim Investigational Site, Kassel
  - 205.452.49105 Boehringer Ingelheim Investigational Site, Kaufbeuren
  - 205.452.49047 Boehringer Ingelheim Investigational Site, Käbschütztal-Krögis
  - 205.452.49101 Boehringer Ingelheim Investigational Site, Koblenz
  - 205.452.49114 Boehringer Ingelheim Investigational Site, Landsberg am Lech
  - 205.452.49169 Boehringer Ingelheim Investigational Site, Langen
  - 205.452.49017 Boehringer Ingelheim Investigational Site, Leipzig
  - 205.452.49035 Boehringer Ingelheim Investigational Site, Leipzig
  - 205.452.49113 Boehringer Ingelheim Investigational Site, Leipzig
  - 205.452.49139 Boehringer Ingelheim Investigational Site, Leipzig
  - 205.452.49172 Boehringer Ingelheim Investigational Site, Leipzig
  - 205.452.49110 Boehringer Ingelheim Investigational Site, Leonberg
  - 205.452.49088 Boehringer Ingelheim Investigational Site, Mannheim
  - 205.452.49108 Boehringer Ingelheim Investigational Site, Marburg
  - 205.452.49122 Boehringer Ingelheim Investigational Site, Marburg
  - 205.452.49055 Boehringer Ingelheim Investigational Site, Minden
  - 205.452.49025 Boehringer Ingelheim Investigational Site, München
  - 205.452.49131 Boehringer Ingelheim Investigational Site, München
  - 205.452.49023 Boehringer Ingelheim Investigational Site, Neumünster
  - 205.452.49132 Boehringer Ingelheim Investigational Site, Neuruppin
  - 205.452.49045 Boehringer Ingelheim Investigational Site, Neuwied
  - 205.452.49062 Boehringer Ingelheim Investigational Site, Oranienburg
  - 205.452.49124 Boehringer Ingelheim Investigational Site, Oschersleben
  - 205.452.49019 Boehringer Ingelheim Investigational Site, Paderborn
  - 205.452.49053 Boehringer Ingelheim Investigational Site, Potsdam
  - 205.452.49076 Boehringer Ingelheim Investigational Site, Potsdam
  - 205.452.49049 Boehringer Ingelheim Investigational Site, Radebeul
  - 205.452.49056 Boehringer Ingelheim Investigational Site, Rathenow
  - 205.452.49009 Boehringer Ingelheim Investigational Site, Raubach
  - 205.452.49002 Boehringer Ingelheim Investigational Site, Rehau
  - 205.452.49142 Boehringer Ingelheim Investigational Site, Reinfeld
  - 205.452.49030 Boehringer Ingelheim Investigational Site, Rhaunen
  - 205.452.49184 Boehringer Ingelheim Investigational Site, Rheine
  - 205.452.49077 Boehringer Ingelheim Investigational Site, Rodgau-Dudenhofen
  - 205.452.49021 Boehringer Ingelheim Investigational Site, Rüsselsheim am Main
  - 205.452.49091 Boehringer Ingelheim Investigational Site, Rüsselsheim am Main
  - 205.452.49042 Boehringer Ingelheim Investigational Site, Saarlouis
  - 205.452.49034 Boehringer Ingelheim Investigational Site, Schwetzingen
  - 205.452.49013 Boehringer Ingelheim Investigational Site, Solingen
  - 205.452.49057 Boehringer Ingelheim Investigational Site, Solingen
  - 205.452.49078 Boehringer Ingelheim Investigational Site, Tübingen
  - 205.452.49099 Boehringer Ingelheim Investigational Site, Ulm
  - 205.452.49043 Boehringer Ingelheim Investigational Site, Wallerfing
  - 205.452.49067 Boehringer Ingelheim Investigational Site, Wardenburg
  - 205.452.49165 Boehringer Ingelheim Investigational Site, Warendorf
  - 205.452.49051 Boehringer Ingelheim Investigational Site, Weinheim
  - 205.452.49127 Boehringer Ingelheim Investigational Site, Weyhe
  - 205.452.49092 Boehringer Ingelheim Investigational Site, Wiesloch
  - 205.452.49018 Boehringer Ingelheim Investigational Site, Witten
  - 205.452.49029 Boehringer Ingelheim Investigational Site, Witten
  - 205.452.49095 Boehringer Ingelheim Investigational Site, Wolfsburg
  - 205.452.49060 Boehringer Ingelheim Investigational Site, Zerbst
- Greece (12):
  - 205.452.30002 Boehringer Ingelheim Investigational Site, Athens
  - 205.452.30003 Boehringer Ingelheim Investigational Site, Athens
  - 205.452.30008 Boehringer Ingelheim Investigational Site, Athens
  - 205.452.30001 Boehringer Ingelheim Investigational Site, Heraklion
  - 205.452.30007 Boehringer Ingelheim Investigational Site, Kalamaria
  - 205.452.30010 Boehringer Ingelheim Investigational Site, Kavala
  - 205.452.30012 Boehringer Ingelheim Investigational Site, Lamia
  - 205.452.30005 Boehringer Ingelheim Investigational Site, Nafplion
  - 205.452.30011 Boehringer Ingelheim Investigational Site, Rethymno
  - 205.452.30006 Boehringer Ingelheim Investigational Site, Serres
  - 205.452.30004 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 205.452.30009 Boehringer Ingelheim Investigational Site, Thessaloniki
- Guatemala (7):
  - 205.452.50205 Boehringer Ingelheim Investigational Site, Guatemala City
  - 205.452.50206 Boehringer Ingelheim Investigational Site, Guatemala City
  - 205.452.50203 Boehringer Ingelheim Investigational Site, Nivel 12
  - 205.452.50201 Boehringer Ingelheim Investigational Site, Nivel Guatemala
  - 205.452.50202 Boehringer Ingelheim Investigational Site, Nivel Guatemala
  - 205.452.50204 Boehringer Ingelheim Investigational Site, Nivel Guatemala
  - 205.452.50207 Boehringer Ingelheim Investigational Site, Quetzaltenango
- Hungary (30):
  - 205.452.36005 Boehringer Ingelheim Investigational Site, Baja
  - 205.452.36004 Boehringer Ingelheim Investigational Site, Budapest
  - 205.452.36016 Boehringer Ingelheim Investigational Site, Budapest
  - 205.452.36030 Boehringer Ingelheim Investigational Site, Budapest
  - 205.452.36007 Boehringer Ingelheim Investigational Site, Debrecen
  - 205.452.36013 Boehringer Ingelheim Investigational Site, Debrecen
  - 205.452.36015 Boehringer Ingelheim Investigational Site, Debrecen
  - 205.452.36029 Boehringer Ingelheim Investigational Site, Deszk
  - 205.452.36026 Boehringer Ingelheim Investigational Site, Dombóvár
  - 205.452.36003 Boehringer Ingelheim Investigational Site, Érd
  - 205.452.36008 Boehringer Ingelheim Investigational Site, Farkasgyepü
  - 205.452.36020 Boehringer Ingelheim Investigational Site, Győr
  - 205.452.36012 Boehringer Ingelheim Investigational Site, Hajduböszörmeny
  - 205.452.36023 Boehringer Ingelheim Investigational Site, Hódmezővásárhely
  - 205.452.36010 Boehringer Ingelheim Investigational Site, Kaposvár
  - 205.452.36018 Boehringer Ingelheim Investigational Site, Kapuvár
  - 205.452.36002 Boehringer Ingelheim Investigational Site, Kecskemét
  - 205.452.36001 Boehringer Ingelheim Investigational Site, Makó
  - 205.452.36006 Boehringer Ingelheim Investigational Site, Mohács
  - 205.452.36022 Boehringer Ingelheim Investigational Site, Mosonmagyaróvár
  - 205.452.36027 Boehringer Ingelheim Investigational Site, Nagykanizsa
  - 205.452.36014 Boehringer Ingelheim Investigational Site, Nyíregyháza
  - 205.452.36009 Boehringer Ingelheim Investigational Site, Pécs
  - 205.452.36011 Boehringer Ingelheim Investigational Site, Pécs
  - 205.452.36028 Boehringer Ingelheim Investigational Site, Siófok
  - 205.452.36021 Boehringer Ingelheim Investigational Site, Szarvas
  - 205.452.36017 Boehringer Ingelheim Investigational Site, Szeged
  - 205.452.36024 Boehringer Ingelheim Investigational Site, Tatabánya
  - 205.452.36019 Boehringer Ingelheim Investigational Site, Törökbálint
  - 205.452.36025 Boehringer Ingelheim Investigational Site, Törökbálint
- India (15):
  - 205.452.91017 Boehringer Ingelheim Investigational Site, Ahmedabad
  - 205.452.91018 Boehringer Ingelheim Investigational Site, Chennai
  - 205.452.91001 Boehringer Ingelheim Investigational Site, Coimbatore
  - 205.452.91002 Boehringer Ingelheim Investigational Site, Coimbatore
  - 205.452.91014 Boehringer Ingelheim Investigational Site, Dadar(East)
  - 205.452.91005 Boehringer Ingelheim Investigational Site, Hyderabad
  - 205.452.91009 Boehringer Ingelheim Investigational Site, Hyderabad
  - 205.452.91004 Boehringer Ingelheim Investigational Site, Jaipur
  - 205.452.91007 Boehringer Ingelheim Investigational Site, Jaipur
  - 205.452.91015 Boehringer Ingelheim Investigational Site, Jaipur
  - 205.452.91016 Boehringer Ingelheim Investigational Site, Jaipur
  - 205.452.91008 Boehringer Ingelheim Investigational Site, Karnataka
  - 205.452.91006 Boehringer Ingelheim Investigational Site, Maharashtra
  - 205.452.91003 Boehringer Ingelheim Investigational Site, Maharastra
  - 205.452.91011 Boehringer Ingelheim Investigational Site, Punjab
- Ireland (8):
  - 205.452.35307 Boehringer Ingelheim Investigational Site, Co. Cork
  - 205.452.35306 Boehringer Ingelheim Investigational Site, Co. Tipperary
  - 205.452.35305 Boehringer Ingelheim Investigational Site, Co. Wexford
  - 205.452.35301 Boehringer Ingelheim Investigational Site, Dublin
  - 205.452.35302 Boehringer Ingelheim Investigational Site, Dublin
  - 205.452.35303 Boehringer Ingelheim Investigational Site, Limerick
  - 205.452.35308 Boehringer Ingelheim Investigational Site, Limerick
  - 205.452.35304 Boehringer Ingelheim Investigational Site, Offaly
- Israel (8):
  - 205.452.97207 Boehringer Ingelheim Investigational Site, Ashkelon
  - 205.452.97204 Boehringer Ingelheim Investigational Site, Beersheba
  - 205.452.97208 Boehringer Ingelheim Investigational Site, Haifa
  - 205.452.97202 Boehringer Ingelheim Investigational Site, Jerusalem
  - 205.452.97206 Boehringer Ingelheim Investigational Site, Kfar Saba
  - 205.452.97203 Boehringer Ingelheim Investigational Site, Petah Tikva
  - 205.452.97201 Boehringer Ingelheim Investigational Site, Rehovot
  - 205.452.97205 Boehringer Ingelheim Investigational Site, Tel Aviv
- Italy (25):
  - 205.452.39003 Boehringer Ingelheim Investigational Site, Arenzano (ge)
  - 205.452.39019 Boehringer Ingelheim Investigational Site, Ascoli Piceno
  - 205.452.39016 Boehringer Ingelheim Investigational Site, Avellino
  - 205.452.39007 Boehringer Ingelheim Investigational Site, Benevento
  - 205.452.39024 Boehringer Ingelheim Investigational Site, Brescia
  - 205.452.39029 Boehringer Ingelheim Investigational Site, Busto Arsizio (va)
  - 205.452.39011 Boehringer Ingelheim Investigational Site, Cagliari
  - 205.452.39013 Boehringer Ingelheim Investigational Site, Cagliari
  - 205.452.39020 Boehringer Ingelheim Investigational Site, Cagliari
  - 205.452.39015 Boehringer Ingelheim Investigational Site, Catanzaro
  - 205.452.39006 Boehringer Ingelheim Investigational Site, Chieti Scalo
  - 205.452.39001 Boehringer Ingelheim Investigational Site, Florence
  - 205.452.39021 Boehringer Ingelheim Investigational Site, Monza
  - 205.452.39014 Boehringer Ingelheim Investigational Site, Napoli
  - 205.452.39012 Boehringer Ingelheim Investigational Site, Orbassano (to)
  - 205.452.39026 Boehringer Ingelheim Investigational Site, Orbassano (to)
  - 205.452.39010 Boehringer Ingelheim Investigational Site, Palermo
  - 205.452.39005 Boehringer Ingelheim Investigational Site, Parma
  - 205.452.39009 Boehringer Ingelheim Investigational Site, Perugia
  - 205.452.39002 Boehringer Ingelheim Investigational Site, Prato
  - 205.452.39030 Boehringer Ingelheim Investigational Site, Reggio Emilia
  - 205.452.39004 Boehringer Ingelheim Investigational Site, Roma
  - 205.452.39017 Boehringer Ingelheim Investigational Site, Roma
  - 205.452.39027 Boehringer Ingelheim Investigational Site, Roma
  - 205.452.39023 Boehringer Ingelheim Investigational Site, Treviso
- Latvia (10):
  - 205.452.37106 Boehringer Ingelheim Investigational Site, Daugavpils
  - 205.452.37107 Boehringer Ingelheim Investigational Site, Daugavpils
  - 205.452.37108 Boehringer Ingelheim Investigational Site, Daugavpils
  - 205.452.37102 Boehringer Ingelheim Investigational Site, Krāslava
  - 205.452.37104 Boehringer Ingelheim Investigational Site, Riga
  - 205.452.37105 Boehringer Ingelheim Investigational Site, Riga
  - 205.452.37109 Boehringer Ingelheim Investigational Site, Riga
  - 205.452.37110 Boehringer Ingelheim Investigational Site, Riga
  - 205.452.37101 Boehringer Ingelheim Investigational Site, Talsi
  - 205.452.37103 Boehringer Ingelheim Investigational Site, Valmiera
- Lithuania (9):
  - 205.452.37003 Boehringer Ingelheim Investigational Site, Alytus
  - 205.452.37001 Boehringer Ingelheim Investigational Site, Kaunas
  - 205.452.37002 Boehringer Ingelheim Investigational Site, Kaunas
  - 205.452.37005 Boehringer Ingelheim Investigational Site, Klaipėda
  - 205.452.37007 Boehringer Ingelheim Investigational Site, Šiauliai
  - 205.452.37011 Boehringer Ingelheim Investigational Site, Utena
  - 205.452.37004 Boehringer Ingelheim Investigational Site, Vilnius
  - 205.452.37008 Boehringer Ingelheim Investigational Site, Vilnius
  - 205.452.37010 Boehringer Ingelheim Investigational Site, Vilnius
- Malaysia (8):
  - 205.452.60006 Boehringer Ingelheim Investigational Site, Johor Bahru
  - 205.452.60001 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 205.452.60002 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 205.452.60004 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 205.452.60008 Boehringer Ingelheim Investigational Site, Kuala Pahang
  - 205.452.60009 Boehringer Ingelheim Investigational Site, Kuala Selangor
  - 205.452.60005 Boehringer Ingelheim Investigational Site, Sarawak
  - 205.452.60007 Boehringer Ingelheim Investigational Site, Terengganu
- Mexico (6):
  - 205.452.52004 Boehringer Ingelheim Investigational Site, Aguascalientes
  - 205.452.52007 Boehringer Ingelheim Investigational Site, Distrito Federal
  - 205.452.52005 Boehringer Ingelheim Investigational Site, Guadalajara
  - 205.452.52001 Boehringer Ingelheim Investigational Site, México
  - 205.452.52002 Boehringer Ingelheim Investigational Site, Monte Rey
  - 205.452.52003 Boehringer Ingelheim Investigational Site, Zona Río
- Netherlands (9):
  - 205.452.31001 Boehringer Ingelheim Investigational Site, Almere Stad
  - 205.452.31008 Boehringer Ingelheim Investigational Site, Andijk
  - 205.452.31002 Boehringer Ingelheim Investigational Site, Beek
  - 205.452.31012 Boehringer Ingelheim Investigational Site, Beek en Donk
  - 205.452.31003 Boehringer Ingelheim Investigational Site, Ermelo
  - 205.452.31010 Boehringer Ingelheim Investigational Site, Hoogwoud
  - 205.452.31011 Boehringer Ingelheim Investigational Site, Nijverdal
  - 205.452.31007 Boehringer Ingelheim Investigational Site, Oude Pekela
  - 205.452.31005 Boehringer Ingelheim Investigational Site, Roelofarendsveen
- New Zealand (4):
  - 205.452.64004 Boehringer Ingelheim Investigational Site, Christchurch
  - 205.452.64003 Boehringer Ingelheim Investigational Site, Dunedin
  - 205.452.64002 Boehringer Ingelheim Investigational Site, Newtown Wellington NZ
  - 205.452.64001 Boehringer Ingelheim Investigational Site, Tauranga
- Norway (12):
  - 205.452.47008 Boehringer Ingelheim Investigational Site, Drammen
  - 205.452.47009 Boehringer Ingelheim Investigational Site, Fredrikstad
  - 205.452.47001 Boehringer Ingelheim Investigational Site, Hønefoss
  - 205.452.47010 Boehringer Ingelheim Investigational Site, Kløfta
  - 205.452.47007 Boehringer Ingelheim Investigational Site, Kolbjørnsvik
  - 205.452.47005 Boehringer Ingelheim Investigational Site, Løvenstad
  - 205.452.47002 Boehringer Ingelheim Investigational Site, Oslo
  - 205.452.47003 Boehringer Ingelheim Investigational Site, Oslo
  - 205.452.47011 Boehringer Ingelheim Investigational Site, Oslo
  - 205.452.47012 Boehringer Ingelheim Investigational Site, Sandvika
  - 205.452.47004 Boehringer Ingelheim Investigational Site, Svelvik
  - 205.452.47006 Boehringer Ingelheim Investigational Site, Trollåsen
- Panama (3):
  - 205.452.50703 Boehringer Ingelheim Investigational Site, Carrasquilla
  - 205.452.50701 Boehringer Ingelheim Investigational Site, Marbella
  - 205.452.50702 Boehringer Ingelheim Investigational Site, Marbella
- Peru (7):
  - 205.452.51002 Boehringer Ingelheim Investigational Site, Bellavista
  - 205.452.51003 Boehringer Ingelheim Investigational Site, Cusco
  - 205.452.51004 Boehringer Ingelheim Investigational Site, Jesús Maria
  - 205.452.51007 Boehringer Ingelheim Investigational Site, Jesús María
  - 205.452.51005 Boehringer Ingelheim Investigational Site, Lima
  - 205.452.51001 Boehringer Ingelheim Investigational Site, San Isidro
  - 205.452.51006 Boehringer Ingelheim Investigational Site, San Martín de Porres
- Philippines (8):
  - 205.452.63004 Boehringer Ingelheim Investigational Site, Cavite City
  - 205.452.63002 Boehringer Ingelheim Investigational Site, Davao City
  - 205.452.63003 Boehringer Ingelheim Investigational Site, Iloilo City
  - 205.452.63006 Boehringer Ingelheim Investigational Site, Iloilo City
  - 205.452.63001 Boehringer Ingelheim Investigational Site, Manila
  - 205.452.63008 Boehringer Ingelheim Investigational Site, Manila
  - 205.452.63005 Boehringer Ingelheim Investigational Site, Quezon City
  - 205.452.63007 Boehringer Ingelheim Investigational Site, Quezon City
- Poland (47):
  - 205.452.48031 Boehringer Ingelheim Investigational Site, Babice
  - 205.452.48003 Boehringer Ingelheim Investigational Site, Bialystok
  - 205.452.48011 Boehringer Ingelheim Investigational Site, Bialystok
  - 205.452.48014 Boehringer Ingelheim Investigational Site, Bydgoszcz
  - 205.452.48008 Boehringer Ingelheim Investigational Site, Chęciny
  - 205.452.48016 Boehringer Ingelheim Investigational Site, Gdansk
  - 205.452.48019 Boehringer Ingelheim Investigational Site, Gdynia
  - 205.452.48037 Boehringer Ingelheim Investigational Site, Gorzow Wlkp
  - 205.452.48015 Boehringer Ingelheim Investigational Site, Iława
  - 205.452.48033 Boehringer Ingelheim Investigational Site, Katowice
  - 205.452.48039 Boehringer Ingelheim Investigational Site, Katowice
  - 205.452.48044 Boehringer Ingelheim Investigational Site, Katowice
  - 205.452.48009 Boehringer Ingelheim Investigational Site, Krakow
  - 205.452.48021 Boehringer Ingelheim Investigational Site, Krakow
  - 205.452.48029 Boehringer Ingelheim Investigational Site, Krakow
  - 205.452.48030 Boehringer Ingelheim Investigational Site, Krakow
  - 205.452.48048 Boehringer Ingelheim Investigational Site, Krakow
  - 205.452.48043 Boehringer Ingelheim Investigational Site, Libiąż
  - 205.452.48002 Boehringer Ingelheim Investigational Site, Lodz
  - 205.452.48051 Boehringer Ingelheim Investigational Site, Lodz
  - 205.452.48056 Boehringer Ingelheim Investigational Site, Lodz
  - 205.452.48059 Boehringer Ingelheim Investigational Site, Lodz
  - 205.452.48018 Boehringer Ingelheim Investigational Site, Olsztyn
  - 205.452.48025 Boehringer Ingelheim Investigational Site, Ostrow Wielkopolska
  - 205.452.48012 Boehringer Ingelheim Investigational Site, Piaseczno
  - 205.452.48040 Boehringer Ingelheim Investigational Site, Piaseczno
  - 205.452.48026 Boehringer Ingelheim Investigational Site, Poznan
  - 205.452.48027 Boehringer Ingelheim Investigational Site, Poznan
  - 205.452.48058 Boehringer Ingelheim Investigational Site, Poznan
  - 205.452.48060 Boehringer Ingelheim Investigational Site, Rokietnica
  - 205.452.48001 Boehringer Ingelheim Investigational Site, Skierniewice
  - 205.452.48036 Boehringer Ingelheim Investigational Site, Szczecin
  - 205.452.48032 Boehringer Ingelheim Investigational Site, Sławków
  - 205.452.48045 Boehringer Ingelheim Investigational Site, Tarnów
  - 205.452.48057 Boehringer Ingelheim Investigational Site, Tczew
  - 205.452.48004 Boehringer Ingelheim Investigational Site, Torun
  - 205.452.48007 Boehringer Ingelheim Investigational Site, Tranow
  - 205.452.48053 Boehringer Ingelheim Investigational Site, Turek
  - 205.452.48034 Boehringer Ingelheim Investigational Site, Warsaw
  - 205.452.48042 Boehringer Ingelheim Investigational Site, Warsaw
  - 205.452.48049 Boehringer Ingelheim Investigational Site, Warsaw
  - 205.452.48017 Boehringer Ingelheim Investigational Site, Wołomin
  - 205.452.48006 Boehringer Ingelheim Investigational Site, Wroclaw
  - 205.452.48028 Boehringer Ingelheim Investigational Site, Wroclaw
  - 205.452.48035 Boehringer Ingelheim Investigational Site, Wroclaw
  - 205.452.48038 Boehringer Ingelheim Investigational Site, Wroclaw
  - 205.452.48022 Boehringer Ingelheim Investigational Site, Zakopane
- Portugal (8):
  - 205.452.35103 Boehringer Ingelheim Investigational Site, Amadora
  - 205.452.35102 Boehringer Ingelheim Investigational Site, Coimbra
  - 205.452.35107 Boehringer Ingelheim Investigational Site, Lisbon
  - 205.452.35108 Boehringer Ingelheim Investigational Site, Lisbon
  - 205.452.35101 Boehringer Ingelheim Investigational Site, Matosinhos Municipality
  - 205.452.35105 Boehringer Ingelheim Investigational Site, Penafiel
  - 205.452.35106 Boehringer Ingelheim Investigational Site, Vila Nova de Gaia
  - 205.452.35104 Boehringer Ingelheim Investigational Site, Viseu
- Puerto Rico (2):
  - 205.452.01177 Boehringer Ingelheim Investigational Site, Ponce
  - 205.452.01162 Boehringer Ingelheim Investigational Site, San Juan
- Romania (11):
  - 205.452.40008 Boehringer Ingelheim Investigational Site, Brasov
  - 205.452.40012 Boehringer Ingelheim Investigational Site, Brasov
  - 205.452.40001 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.452.40002 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.452.40003 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.452.40004 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.452.40007 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.452.40009 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.452.40013 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.452.40011 Boehringer Ingelheim Investigational Site, Constanța
  - 205.452.40006 Boehringer Ingelheim Investigational Site, Craiova
- Russia (56):
  - 205.452.07030 Boehringer Ingelheim Investigational Site, Arkhangelsk
  - 205.452.07049 Boehringer Ingelheim Investigational Site, Barnaul
  - 205.452.07054 Boehringer Ingelheim Investigational Site, Barnaul
  - 205.452.07053 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 205.452.07038 Boehringer Ingelheim Investigational Site, Gatchina (Leningradskaya Oblast)
  - 205.452.07036 Boehringer Ingelheim Investigational Site, Irkutsk
  - 205.452.07001 Boehringer Ingelheim Investigational Site, Ivanovo
  - 205.452.07023 Boehringer Ingelheim Investigational Site, Kaliningrad
  - 205.452.07003 Boehringer Ingelheim Investigational Site, Kazan'
  - 205.452.07005 Boehringer Ingelheim Investigational Site, Kazan'
  - 205.452.07007 Boehringer Ingelheim Investigational Site, Kazan'
  - 205.452.07048 Boehringer Ingelheim Investigational Site, Kemerovo
  - 205.452.07060 Boehringer Ingelheim Investigational Site, Kemerovo
  - 205.452.07059 Boehringer Ingelheim Investigational Site, Kirov
  - 205.452.07009 Boehringer Ingelheim Investigational Site, Krasnodar
  - 205.452.07010 Boehringer Ingelheim Investigational Site, Krasnodar
  - 205.452.07013 Boehringer Ingelheim Investigational Site, Moscow
  - 205.452.07020 Boehringer Ingelheim Investigational Site, Moscow
  - 205.452.07021 Boehringer Ingelheim Investigational Site, Moscow
  - 205.452.07026 Boehringer Ingelheim Investigational Site, Moscow
  - 205.452.07027 Boehringer Ingelheim Investigational Site, Moscow
  - 205.452.07028 Boehringer Ingelheim Investigational Site, Moscow
  - 205.452.07029 Boehringer Ingelheim Investigational Site, Moscow
  - 205.452.07043 Boehringer Ingelheim Investigational Site, Moscow
  - 205.452.07045 Boehringer Ingelheim Investigational Site, Moscow
  - 205.452.07004 Boehringer Ingelheim Investigational Site, Murmansk
  - 205.452.07051 Boehringer Ingelheim Investigational Site, Nizhny Novgorod
  - 205.452.07055 Boehringer Ingelheim Investigational Site, Nizhny Novgorod
  - 205.452.07037 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 205.452.07040 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 205.452.07042 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 205.452.07041 Boehringer Ingelheim Investigational Site, Penza
  - 205.452.07050 Boehringer Ingelheim Investigational Site, Pskov
  - 205.452.07015 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 205.452.07016 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 205.452.07039 Boehringer Ingelheim Investigational Site, Ryazan
  - 205.452.07002 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.452.07006 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.452.07011 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.452.07014 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.452.07017 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.452.07018 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.452.07022 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.452.07024 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.452.07025 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.452.07033 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.452.07046 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.452.07052 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.452.07034 Boehringer Ingelheim Investigational Site, Samara
  - 205.452.07047 Boehringer Ingelheim Investigational Site, Saratov
  - 205.452.07032 Boehringer Ingelheim Investigational Site, Tomsk
  - 205.452.07035 Boehringer Ingelheim Investigational Site, Tomsk
  - 205.452.07057 Boehringer Ingelheim Investigational Site, Tomsk
  - 205.452.07019 Boehringer Ingelheim Investigational Site, Veliky Novgorod
  - 205.452.07044 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 205.452.07031 Boehringer Ingelheim Investigational Site, Yekaterinburg
- Serbia (7):
  - 205.452.38103 Boehringer Ingelheim Investigational Site, Belgrade
  - 205.452.38104 Boehringer Ingelheim Investigational Site, Belgrade
  - 205.452.38106 Boehringer Ingelheim Investigational Site, Belgrade
  - 205.452.38107 Boehringer Ingelheim Investigational Site, Belgrade
  - 205.452.38101 Boehringer Ingelheim Investigational Site, Kamenitz
  - 205.452.38102 Boehringer Ingelheim Investigational Site, Kragujevac
  - 205.452.38105 Boehringer Ingelheim Investigational Site, Niš
- Slovakia (13):
  - 205.452.42103 Boehringer Ingelheim Investigational Site, Bardejov
  - 205.452.42107 Boehringer Ingelheim Investigational Site, Bratislava
  - 205.452.42102 Boehringer Ingelheim Investigational Site, Humenné
  - 205.452.42105 Boehringer Ingelheim Investigational Site, Košice
  - 205.452.42111 Boehringer Ingelheim Investigational Site, Košice
  - 205.452.42113 Boehringer Ingelheim Investigational Site, Košice
  - 205.452.42108 Boehringer Ingelheim Investigational Site, Levice
  - 205.452.42109 Boehringer Ingelheim Investigational Site, Martin
  - 205.452.42112 Boehringer Ingelheim Investigational Site, Poprad
  - 205.452.42101 Boehringer Ingelheim Investigational Site, Prešov
  - 205.452.42104 Boehringer Ingelheim Investigational Site, Rimavská Sobota
  - 205.452.42106 Boehringer Ingelheim Investigational Site, Spišská Nová Ves
  - 205.452.42110 Boehringer Ingelheim Investigational Site, Štúrovo
- South Africa (14):
  - 205.452.27002 Boehringer Ingelheim Investigational Site, Bellville
  - 205.452.27010 Boehringer Ingelheim Investigational Site, Bloemfontein
  - 205.452.27001 Boehringer Ingelheim Investigational Site, Cape Town
  - 205.452.27004 Boehringer Ingelheim Investigational Site, Cape Town
  - 205.452.27008 Boehringer Ingelheim Investigational Site, Cape Town
  - 205.452.27011 Boehringer Ingelheim Investigational Site, Cape Town
  - 205.452.27012 Boehringer Ingelheim Investigational Site, Cape Town
  - 205.452.27006 Boehringer Ingelheim Investigational Site, Centurion
  - 205.452.27003 Boehringer Ingelheim Investigational Site, Durban
  - 205.452.27013 Boehringer Ingelheim Investigational Site, eManzimtoti
  - 205.452.27014 Boehringer Ingelheim Investigational Site, Johannesburg
  - 205.452.27005 Boehringer Ingelheim Investigational Site, Pretoria
  - 205.452.27009 Boehringer Ingelheim Investigational Site, Pretoria
  - 205.452.27007 Boehringer Ingelheim Investigational Site, Somerset West
- South Korea (20):
  - 205.452.82008 Boehringer Ingelheim Investigational Site, Bucheon-si
  - 205.452.82002 Boehringer Ingelheim Investigational Site, Busan
  - 205.452.82012 Boehringer Ingelheim Investigational Site, Busan
  - 205.452.82010 Boehringer Ingelheim Investigational Site, Daegu
  - 205.452.82016 Boehringer Ingelheim Investigational Site, Daejoen
  - 205.452.82009 Boehringer Ingelheim Investigational Site, Gangwon-Do
  - 205.452.82017 Boehringer Ingelheim Investigational Site, Goyang
  - 205.452.82004 Boehringer Ingelheim Investigational Site, Gwangju
  - 205.452.82005 Boehringer Ingelheim Investigational Site, Incheon
  - 205.452.82020 Boehringer Ingelheim Investigational Site, Jeonju
  - 205.452.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 205.452.82003 Boehringer Ingelheim Investigational Site, Seoul
  - 205.452.82006 Boehringer Ingelheim Investigational Site, Seoul
  - 205.452.82007 Boehringer Ingelheim Investigational Site, Seoul
  - 205.452.82011 Boehringer Ingelheim Investigational Site, Seoul
  - 205.452.82013 Boehringer Ingelheim Investigational Site, Seoul
  - 205.452.82014 Boehringer Ingelheim Investigational Site, Seoul
  - 205.452.82015 Boehringer Ingelheim Investigational Site, Seoul
  - 205.452.82018 Boehringer Ingelheim Investigational Site, Seoul
  - 205.452.82019 Boehringer Ingelheim Investigational Site, Uijeongbu-si
- Spain (24):
  - 205.452.34018 Boehringer Ingelheim Investigational Site, Badajoz
  - 205.452.34021 Boehringer Ingelheim Investigational Site, Badalona (Barcelona)
  - 205.452.34010 Boehringer Ingelheim Investigational Site, Barcelona
  - 205.452.34025 Boehringer Ingelheim Investigational Site, Barcelona
  - 205.452.34015 Boehringer Ingelheim Investigational Site, Cáceres
  - 205.452.34027 Boehringer Ingelheim Investigational Site, Centelles
  - 205.452.34016 Boehringer Ingelheim Investigational Site, Elda
  - 205.452.34008 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 205.452.34026 Boehringer Ingelheim Investigational Site, Lugo
  - 205.452.34011 Boehringer Ingelheim Investigational Site, Madrid
  - 205.452.34019 Boehringer Ingelheim Investigational Site, Madrid
  - 205.452.34020 Boehringer Ingelheim Investigational Site, Málaga
  - 205.452.34002 Boehringer Ingelheim Investigational Site, Mérida
  - 205.452.34017 Boehringer Ingelheim Investigational Site, Plasencia
  - 205.452.34001 Boehringer Ingelheim Investigational Site, Pozuelo de Alarcón
  - 205.452.34024 Boehringer Ingelheim Investigational Site, Sant Joan d'Alacant
  - 205.452.34003 Boehringer Ingelheim Investigational Site, Santander
  - 205.452.34005 Boehringer Ingelheim Investigational Site, Terrassa (Barcelona)
  - 205.452.34007 Boehringer Ingelheim Investigational Site, Torrevieja
  - 205.452.34012 Boehringer Ingelheim Investigational Site, Valencia
  - 205.452.34013 Boehringer Ingelheim Investigational Site, Valladolid
  - 205.452.34009 Boehringer Ingelheim Investigational Site, Vic (Barcelona)
  - 205.452.34023 Boehringer Ingelheim Investigational Site, Vilanova i la Geltrú
  - 205.452.34004 Boehringer Ingelheim Investigational Site, Zaragoza
- Sweden (13):
  - 205.452.46005 Boehringer Ingelheim Investigational Site, Brämhult
  - 205.452.46014 Boehringer Ingelheim Investigational Site, Eksjö
  - 205.452.46013 Boehringer Ingelheim Investigational Site, Gothenburg
  - 205.452.46012 Boehringer Ingelheim Investigational Site, Gullspång
  - 205.452.46001 Boehringer Ingelheim Investigational Site, Höllviken
  - 205.452.46008 Boehringer Ingelheim Investigational Site, Järfälla
  - 205.452.46009 Boehringer Ingelheim Investigational Site, Kil
  - 205.452.46007 Boehringer Ingelheim Investigational Site, Lidingö
  - 205.452.46003 Boehringer Ingelheim Investigational Site, Luleå
  - 205.452.46006 Boehringer Ingelheim Investigational Site, Örebro
  - 205.452.46010 Boehringer Ingelheim Investigational Site, Sigtuna
  - 205.452.46002 Boehringer Ingelheim Investigational Site, Solna
  - 205.452.46011 Boehringer Ingelheim Investigational Site, Uddevalla
- Switzerland (13):
  - 205.452.41003 Boehringer Ingelheim Investigational Site, Ascona
  - 205.452.41004 Boehringer Ingelheim Investigational Site, Basel
  - 205.452.41016 Boehringer Ingelheim Investigational Site, Bern
  - 205.452.41012 Boehringer Ingelheim Investigational Site, Glarus
  - 205.452.41001 Boehringer Ingelheim Investigational Site, Gossau
  - 205.452.41015 Boehringer Ingelheim Investigational Site, Liestal
  - 205.452.41010 Boehringer Ingelheim Investigational Site, Locarno
  - 205.452.41011 Boehringer Ingelheim Investigational Site, Lugano
  - 205.452.41002 Boehringer Ingelheim Investigational Site, Sankt Gallen
  - 205.452.41009 Boehringer Ingelheim Investigational Site, Sankt Gallen
  - 205.452.41007 Boehringer Ingelheim Investigational Site, Spiez
  - 205.452.41013 Boehringer Ingelheim Investigational Site, Zurich
  - 205.452.41014 Boehringer Ingelheim Investigational Site, Zurich
- Taiwan (14):
  - 205.452.88607 Boehringer Ingelheim Investigational Site, Changhua
  - 205.452.88614 Boehringer Ingelheim Investigational Site, Chiayi City
  - 205.452.88608 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 205.452.88609 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 205.452.88611 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 205.452.88604 Boehringer Ingelheim Investigational Site, New Taipei City
  - 205.452.88605 Boehringer Ingelheim Investigational Site, Taichung
  - 205.452.88606 Boehringer Ingelheim Investigational Site, Taichung
  - 205.452.88612 Boehringer Ingelheim Investigational Site, Taichung
  - 205.452.88610 Boehringer Ingelheim Investigational Site, Tainan
  - 205.452.88602 Boehringer Ingelheim Investigational Site, Taipei
  - 205.452.88603 Boehringer Ingelheim Investigational Site, Taipei
  - 205.452.88613 Boehringer Ingelheim Investigational Site, Taipei
  - 205.452.88601 Boehringer Ingelheim Investigational Site, Taoyuan
- Thailand (5):
  - 205.452.66004 Boehringer Ingelheim Investigational Site, Chiang Mai
  - 205.452.66003 Boehringer Ingelheim Investigational Site, Hatyai, Songkhla
  - 205.452.66002 Boehringer Ingelheim Investigational Site, Khon Kaen
  - 205.452.66001 Boehringer Ingelheim Investigational Site, Nonthaburi
  - 205.452.66005 Boehringer Ingelheim Investigational Site, Phitsanulok
- Tunisia (10):
  - 205.452.21603 Boehringer Ingelheim Investigational Site, Aryanah
  - 205.452.21605 Boehringer Ingelheim Investigational Site, Aryanah
  - 205.452.21606 Boehringer Ingelheim Investigational Site, Aryanah
  - 205.452.21607 Boehringer Ingelheim Investigational Site, Aryanah
  - 205.452.21610 Boehringer Ingelheim Investigational Site, Mahdia
  - 205.452.21609 Boehringer Ingelheim Investigational Site, Monastir
  - 205.452.21608 Boehringer Ingelheim Investigational Site, Nabeul
  - 205.452.21601 Boehringer Ingelheim Investigational Site, Tunis
  - 205.452.21602 Boehringer Ingelheim Investigational Site, Tunis
  - 205.452.21604 Boehringer Ingelheim Investigational Site, Tunis
- Turkey (Türkiye) (16):
  - 205.452.90001 Boehringer Ingelheim Investigational Site, Adana
  - 205.452.90008 Boehringer Ingelheim Investigational Site, Ankara
  - 205.452.90013 Boehringer Ingelheim Investigational Site, Ankara
  - 205.452.90005 Boehringer Ingelheim Investigational Site, Antalya
  - 205.452.90018 Boehringer Ingelheim Investigational Site, Aydin
  - 205.452.90003 Boehringer Ingelheim Investigational Site, Bolu
  - 205.452.90006 Boehringer Ingelheim Investigational Site, Edirne
  - 205.452.90010 Boehringer Ingelheim Investigational Site, Erzurum
  - 205.452.90019 Boehringer Ingelheim Investigational Site, Hatay
  - 205.452.90017 Boehringer Ingelheim Investigational Site, Istanbul
  - 205.452.90020 Boehringer Ingelheim Investigational Site, Istanbul
  - 205.452.90021 Boehringer Ingelheim Investigational Site, Istanbul
  - 205.452.90015 Boehringer Ingelheim Investigational Site, Izmir
  - 205.452.90016 Boehringer Ingelheim Investigational Site, Izmir
  - 205.452.90022 Boehringer Ingelheim Investigational Site, Izmir
  - 205.452.90007 Boehringer Ingelheim Investigational Site, Malatya
- Ukraine (26):
  - 205.452.38028 Boehringer Ingelheim Investigational Site, Crimea
  - 205.452.38024 Boehringer Ingelheim Investigational Site, Dnipropetrovks
  - 205.452.38022 Boehringer Ingelheim Investigational Site, Dnipropetrovsk
  - 205.452.38034 Boehringer Ingelheim Investigational Site, Dnyepropyetrovsk
  - 205.452.38002 Boehringer Ingelheim Investigational Site, Donetsk
  - 205.452.38020 Boehringer Ingelheim Investigational Site, Donetsk
  - 205.452.38011 Boehringer Ingelheim Investigational Site, Ivano-Frankivsk
  - 205.452.38001 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.452.38004 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.452.38005 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.452.38006 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.452.38008 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.452.38018 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.452.38003 Boehringer Ingelheim Investigational Site, Kiev
  - 205.452.38010 Boehringer Ingelheim Investigational Site, Kiev
  - 205.452.38012 Boehringer Ingelheim Investigational Site, Kiev
  - 205.452.38013 Boehringer Ingelheim Investigational Site, Kiev
  - 205.452.38015 Boehringer Ingelheim Investigational Site, Kiev
  - 205.452.38032 Boehringer Ingelheim Investigational Site, Kiev
  - 205.452.38026 Boehringer Ingelheim Investigational Site, Nikolayev
  - 205.452.38023 Boehringer Ingelheim Investigational Site, Odesa
  - 205.452.38027 Boehringer Ingelheim Investigational Site, Odesa
  - 205.452.38031 Boehringer Ingelheim Investigational Site, Odesa
  - 205.452.38017 Boehringer Ingelheim Investigational Site, Simferopol
  - 205.452.38019 Boehringer Ingelheim Investigational Site, Vinnytsia
  - 205.452.38030 Boehringer Ingelheim Investigational Site, Zaporizhzhya
- United Kingdom (10):
  - 205.452.44010 Boehringer Ingelheim Investigational Site, Atherstone
  - 205.452.44008 Boehringer Ingelheim Investigational Site, Burbage
  - 205.452.44004 Boehringer Ingelheim Investigational Site, Chertsey
  - 205.452.44002 Boehringer Ingelheim Investigational Site, Chesterfield
  - 205.452.44003 Boehringer Ingelheim Investigational Site, Coventry
  - 205.452.44001 Boehringer Ingelheim Investigational Site, Exeter
  - 205.452.44007 Boehringer Ingelheim Investigational Site, Fowey
  - 205.452.44005 Boehringer Ingelheim Investigational Site, Frome
  - 205.452.44011 Boehringer Ingelheim Investigational Site, Royal Leamington Spa
  - 205.452.44006 Boehringer Ingelheim Investigational Site, Saint Just, Penzance

REFERENCES:
- [Derived] Wise RA, Calverley PM, Carter K, Clerisme-Beaty E, Metzdorf N, Anzueto A. Seasonal variations in exacerbations and deaths in patients with COPD during the TIOSPIR(R) trial. Int J Chron Obstruct Pulmon Dis. 2018 Feb 14;13:605-616. doi: 10.2147/COPD.S148393. eCollection 2018. PMID 29497289
- [Derived] Calverley PMA, Mueller A, Fowler A, Metzdorf N, Wise RA. The Effect of Defining Chronic Obstructive Pulmonary Disease by the Lower Limit of Normal of FEV1/FVC Ratio in Tiotropium Safety and Performance in Respimat Participants. Ann Am Thorac Soc. 2018 Feb;15(2):200-208. doi: 10.1513/AnnalsATS.201703-194OC. PMID 28957643
- [Derived] Dahl R, Calverley PM, Anzueto A, Metzdorf N, Fowler A, Mueller A, Wise R, Dusser D. Safety and efficacy of tiotropium in patients switching from HandiHaler to Respimat in the TIOSPIR trial. BMJ Open. 2015 Dec 29;5(12):e009015. doi: 10.1136/bmjopen-2015-009015. PMID 26715479
- [Derived] Anzueto A, Wise R, Calverley P, Dusser D, Tang W, Metzdorf N, Dahl R. The Tiotropium Safety and Performance in Respimat(R) (TIOSPIR(R)) Trial: Spirometry Outcomes. Respir Res. 2015 Sep 15;16(1):107. doi: 10.1186/s12931-015-0269-4. PMID 26369563
- [Derived] Wise RA, Anzueto A, Cotton D, Dahl R, Devins T, Disse B, Dusser D, Joseph E, Kattenbeck S, Koenen-Bergmann M, Pledger G, Calverley P; TIOSPIR Investigators. Tiotropium Respimat inhaler and the risk of death in COPD. N Engl J Med. 2013 Oct 17;369(16):1491-501. doi: 10.1056/NEJMoa1303342. Epub 2013 Aug 30. PMID 23992515

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This table summarizes study treatment disposition and reasons for discontinuation of study medication. Deaths that caused discontinuation from trial medications are included in AEs. Lost to follow-up indicates status at time of discontinuation of trial medication. Vital status was ascertained for 99.7% of patients.
Period: Overall Study
Arm/Group | Tiotropium 2.5 mcg and Placebo | Tiotropium 5 mcg and Placebo | Tiotropium 18 mcg and Placebo
Started | 5741 | 5729 | 5713
Completed | 4400 (See Pre-Assignment Details above for comments.) | 4399 (See Pre-Assignment Details above for comments.) | 4400 (See Pre-Assignment Details above for comments.)
Not Completed | 1341 | 1330 | 1313
Not completed — Not treated | 11 | 18 | 19
Not completed — Sites with data irregularities/fraud | 6 | 6 | 7
Not completed — Adverse Event | 602 | 606 | 635
Not completed — Lack of Efficacy | 65 | 60 | 59
Not completed — Protocol Violation | 64 | 66 | 41
Not completed — Lost to Follow-up | 52 | 63 | 55
Not completed — Withdrawal by Subject | 331 | 335 | 319
Not completed — Other reason not specified | 210 | 176 | 178

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This analysis set included all randomized subjects without data irregularities who were documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium 2.5 mcg and Placebo | Tiotropium 5 mcg and Placebo | Tiotropium 18 mcg and Placebo | Total
Number analyzed (Participants) | 5724 | 5705 | 5687 | 17116
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (9.1) | 64.9 (9.1) | 65.0 (9.0) | 65.0 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1656 | 1571 | 1652 | 4879
  Male | 4068 | 4134 | 4035 | 12237

OUTCOME MEASURES:

1. Primary Outcome: Time to All-Cause Mortality
Description: Number of patients with all-cause mortality
Time Frame: Up to 3 years
Population: Death analysis set (DAS) including vital status follow-up: This analysis set included all randomized subjects excluding only subjects who were documented as not treated.
Measure: Number; unit: Number of deaths
Arm/Group | Tiotropium 2.5 mcg and Placebo | Tiotropium 5 mcg and Placebo | Tiotropium 18 mcg and Placebo
Number analyzed (Participants) | 5730 | 5711 | 5694
Number of deaths | 440 (7.7) | 423 (7.4) | 439 (7.7)
Statistical Analysis 1: Comparison: Tiotropium 5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; H0: Hazard Ratio for Respimat/HandiHaler >= 1.25 Ha: Hazard Ratio for Respimat/HandiHaler < 1.25; Test type: Non-Inferiority or Equivalence — Three tests were conducted in hierarchical order. Non-inferiority of time to death from any cause was tested on the two Respimat doses: Tio R 5 vs. Tio HH18, then if non-inferiority was achieved Tio R 2.5 vs Tio HH18. If successful, a test of superiority of Tio R5 over Tio HH18 for time to first COPD exacerbation was conducted. The non-inferiority delta for time to death was 1.25. Non-inferiority tests were performed at one-sided α=0.025 level. Superiority test was performed at two sided α=0.05; Regression, Cox; Hazard Ratio (HR) = 0.957, 95% CI 2-sided [0.837 to 1.094]
Statistical Analysis 2: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; H0: Hazard Ratio for Respimat/HandiHaler >= 1.25 Ha: Hazard Ratio for Respimat/HandiHaler < 1.25; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Regression, Cox; Hazard Ratio (HR) = 0.996, 95% CI 2-sided [0.872 to 1.136]

2. Primary Outcome: Time to First COPD Exacerbation
Description: Defined as "a complex of lower respiratory events/symptoms (increase of new onset) related to the underlying COPD, with duration of three days or more, requiring a change in treatment" where a "complex of lower respiratory event/symptoms" was defined as having at least two of the following: shortness of breath, sputum production (volume), occurrence of purulent sputum, cough, wheezing, chest tightness and where "a required change in treatment" includes the following:Prescription of antibiotics and/or systemic steroids, and/or a newly prescribed maintenance respiratory medication (i.e., bronchodilators including theophyllines).
  "Onset of exacerbation" was defined by the onset of first recorded symptom. The "end of exacerbation" was decided by the investigator based on clinical judgement.
  Exacerbations were classified as follows:
  Mild:a new prescription of maintenance bronchodilator only Moderate:antibiotics or systemic steroids without hospitalization Severe:hospitalization.
Time Frame: Up to 3 years
Population: Treated set (TS, on-treatment only)
Measure: Median (95% Confidence Interval); unit: days to event
Arm/Group | Tiotropium 2.5 mcg and Placebo | Tiotropium 5 mcg and Placebo | Tiotropium 18 mcg and Placebo
Number analyzed (Participants) | 5724 | 5705 | 5687
days to event | 707 [662 to 750] | 756 [692 to 816] | 719 [672 to 777]
Statistical Analysis 1: Comparison: Tiotropium 5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; H0: Hazard Ratio for Respimat/HandiHaler = 1 Ha: Hazard Ratio for Respimat/HandiHaler ≠ 1 at alpha = 0.05; Test type: Superiority or Other; p = 0.4194, Regression, Cox; Hazard Ratio (HR) = 0.978, 95% CI 2-sided [0.928 to 1.032]
Statistical Analysis 2: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; H0: Hazard Ratio for Respimat/HandiHaler = 1 Ha: Hazard Ratio for Respimat/HandiHaler ≠ 1 at alpha = 0.05; Test type: Superiority or Other; p = 0.5593, Regression, Cox; Hazard Ratio (HR) = 1.016, 95% CI 2-sided [0.964 to 1.070]
Statistical Analysis 3: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 5 mcg and Placebo; H0: Hazard Ratio for Respimat/HandiHaler = 1 Ha: Hazard Ratio for Respimat/HandiHaler ≠ 1 at alpha = 0.05; Test type: Superiority or Other; p = 0.1639, Regression, Cox; Hazard Ratio (HR) = 1.038, 95% CI 2-sided [0.985 to 1.094]

3. Secondary Outcome: Trough FEV1 Over 120 Weeks (in a Substudy of 1370 Patients)
Description: Trough forced expiratory volume in one second (FEV1) over 120 weeks (in a substudy of 1370 patients)
Time Frame: Up to 3 years
Population: SSS - PFT - Sub-study set (pulmonary function testing). This analysis set included all subjects in the TS who signed informed consent to participate in the spirometry sub-study and had at least baseline and one on-treatment trough FEV1.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Tiotropium 2.5 mcg and Placebo | Tiotropium 5 mcg and Placebo | Tiotropium 18 mcg and Placebo
Number analyzed (Participants) | 464 | 461 | 445
Liter | 1.258 (0.012) | 1.285 (0.012) | 1.295 (0.012)
Statistical Analysis 1: Comparison: Tiotropium 5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; FEV1 was analyzed through Week 120 using REML-based repeated measures. H0: Adjusted mean difference for Respimat/HandiHaler ≥ 50ml Ha: Adjusted mean difference for Respimat/HandiHaler < 50 ml; Test type: Non-Inferiority or Equivalence — The first test performed was to test the main effect for treatment in the mixed model repeated measures (MMRM) model, specifically the 95% CI for the contrast between Tio R 5ug and Tio HH 18ug was compared to the non-inferiority delta of 50 mL. If that test was successful, the second test in the hierarchy was to test the main effect for treatment in the MMRM model, specifically the 95% CI for the contrast between Tio R 2.5 ug and Tio HH 18 ug was compared to the non-inferiority delta of 50 mL; Mixed Model Repeated Measures — An autoregression-1 covariance structure modeled the within-subject errors because visits were equally spaced. The Kenward-Roger approximation estimated denominator degrees of freedom; Adjusted mean difference = -.010, 95% CI 2-sided [-.038 to 0.018], Standard Error of Mean 0.014 — Model included the fixed, categorical effects of treatment, investigative site, visit, and treatment-by-visit interaction, and continuous, fixed covariates of baseline and baseline-by-visit interaction, and a random term of patient
Statistical Analysis 2: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mixed Model Repeated Measures — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -.037, 95% CI 2-sided [-.065 to -.009], Standard Error of Mean 0.014 — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Number of COPD Exacerbations
Description: The number of COPD exacerbations. COPD exacerbation defined as "a complex of lower respiratory events/symptoms (increase of new onset) related to the underlying COPD, with duration of three days or more, requiring a change in treatment" where a "complex of lower respiratory event/symptoms" was defined as having at least two of the following: shortness of breath, sputum production (volume), occurrence of purulent sputum, cough, wheezing, chest tightness and where "a required change in treatment" includes the following:Prescription of antibiotics and/or systemic steroids, and/or a newly prescribed maintenance respiratory medication (i.e., bronchodilators including theophyllines).
Time Frame: Up to 3 years
Population: Treated Set - on treatment only
Measure: Number; unit: number of COPD exacerbations
Arm/Group | Tiotropium 2.5 mcg and Placebo | Tiotropium 5 mcg and Placebo | Tiotropium 18 mcg and Placebo
Number analyzed (Participants) | 5724 | 5705 | 5687
number of COPD exacerbations | 6565 | 6425 | 6504
Statistical Analysis 1: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; Test type: Superiority or Other; p = 0.8330, Negative binomial regression; Rate ratio of events = 1.01, 95% CI 2-sided [0.95 to 1.06], Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: Tiotropium 5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; Test type: Superiority or Other; p = 0.8047, Negative binomial regression; Rate ratio of events = 0.99, 95% CI 2-sided [0.94 to 1.05], Standard Error of Mean 0.03
Statistical Analysis 3: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 5 mcg and Placebo; Test type: Superiority or Other; p = 0.6468, Negative binomial regression; Rate ratio of events = 1.01, 95% CI 2-sided [0.96 to 1.07], Standard Error of Mean 0.03

5. Secondary Outcome: Time to First Hospitalization Associated With COPD Exacerbation
Description: The results presented below are for the patients with hospitalizations due to COPD exacerbations.
Time Frame: Up to 3 years
Population: treated set - on-treatment only
Measure: Number; unit: Number of patients with event
Arm/Group | Tiotropium 2.5 mcg and Placebo | Tiotropium 5 mcg and Placebo | Tiotropium 18 mcg and Placebo
Number analyzed (Participants) | 5724 | 5705 | 5687
Number of patients with event | 869 | 826 | 811
Statistical Analysis 1: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; Test type: Superiority or Other; p = 0.1762, Regression, Cox; Hazard Ratio (HR) = 1.068, 95% CI 2-sided [0.971 to 1.176]
Statistical Analysis 2: Comparison: Tiotropium 5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; Test type: Superiority or Other; p = 0.6384, Regression, Cox; Hazard Ratio (HR) = 1.024, 95% CI 2-sided [0.929 to 1.128]
Statistical Analysis 3: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 5 mcg and Placebo; Test type: Superiority or Other; p = 0.3784, Regression, Cox; Hazard Ratio (HR) = 1.044, 95% CI 2-sided [0.949 to 1.148]

6. Secondary Outcome: Number of Hospitalizations Associated With COPD Exacerbation
Description: Total number of hospitalizations associated with COPD exacerbation.
Time Frame: Up to 3 years
Population: treated set - on treatment only
Measure: Number; unit: number of hospitalizations
Arm/Group | Tiotropium 2.5 mcg and Placebo | Tiotropium 5 mcg and Placebo | Tiotropium 18 mcg and Placebo
Number analyzed (Participants) | 5724 | 5705 | 5687
number of hospitalizations | 1316 | 1284 | 1216
Statistical Analysis 1: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; Test type: Superiority or Other; p = 0.1255, Negative binomial regression — p-value from negative binomial regression; Rate ratio of events = 1.09, 95% CI 2-sided [0.98 to 1.22], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Tiotropium 5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; Test type: Superiority or Other; p = 0.3441, Negative binomial regression — p-value from negative binomial regression; Rate ratio of events = 1.06, 95% CI 2-sided [0.94 to 1.18], Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 5 mcg and Placebo; Test type: Superiority or Other; p = 0.5573, Negative binomial regression — p-value from negative binomial regression; Rate ratio of events = 1.03, 95% CI 2-sided [0.92 to 1.16], Standard Error of Mean 0.06

7. Secondary Outcome: Time to First Moderate to Severe COPD Exacerbation
Description: COPD exacerbation defined as "a complex of lower respiratory events/symptoms (increase of new onset) related to the underlying COPD, with duration of three days or more, requiring a change in treatment" where a "complex of lower respiratory event/symptoms" was defined as having at least two of the following: shortness of breath, sputum production (volume), occurrence of purulent sputum, cough, wheezing, chest tightness and where "a required change in treatment" includes the following:Prescription of antibiotics and/or systemic steroids, and/or a newly prescribed maintenance respiratory medication (i.e., bronchodilators including theophyllines).
  Exacerbations classified as follows:
  Mild:a new prescription of maintenance bronchodilator only Moderate:antibiotics or systemic steroids without hospitalization Severe:hospitalization.
  Results presented below are number of patients with moderate to severe exacerbations.
Time Frame: Up to 3 years
Population: treated set - on treatment only
Measure: Number; unit: number of patients with event
Arm/Group | Tiotropium 2.5 mcg and Placebo | Tiotropium 5 mcg and Placebo | Tiotropium 18 mcg and Placebo
Number analyzed (Participants) | 5724 | 5705 | 5687
number of patients with event | 2769 | 2694 | 2732
Statistical Analysis 1: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; Test type: Superiority or Other; p = 0.6823, Regression, Cox; Hazard Ratio (HR) = 1.011, 95% CI 2-sided [0.959 to 1.066]
Statistical Analysis 2: Comparison: Tiotropium 5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; Test type: Superiority or Other; p = 0.5377, Regression, Cox; Hazard Ratio (HR) = 0.983, 95% CI 2-sided [0.932 to 1.037]
Statistical Analysis 3: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 5 mcg and Placebo; Test type: Superiority or Other; p = 0.3048, Regression, Cox; Hazard Ratio (HR) = 1.028, 95% CI 2-sided [0.975 to 1.084]

8. Secondary Outcome: Time to Onset of First Major Adverse Cardiovascular Event (MACE)
Description: Time to onset of first major adverse cardiovascular event (MACE). MACE was defined as: Fatal event in the system organ classes of cardiac and vascular disorders, Preferred terms: sudden death, cardiac death, sudden cardiac death, Outcome events of myocardial infarction (serious and non-serious), Outcome events of stroke (serious and non-serious) and Outcome events of TIA (serious and non-serious). The results presented below are for the number of patients with MACE.
Time Frame: Up to 3 years
Population: Treated set - on treatment only
Measure: Number; unit: number of patients with MACE
Arm/Group | Tiotropium 2.5 mcg and Placebo | Tiotropium 5 mcg and Placebo | Tiotropium 18 mcg and Placebo
Number analyzed (Participants) | 5724 | 5705 | 5687
number of patients with MACE | 224 | 222 | 202
Statistical Analysis 1: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; Causes of death from MACE were determined by adjudication; Test type: Superiority or Other; p = 0.3043, Regression, Cox; Hazard Ratio (HR) = 1.105, 95% CI 2-sided [0.913 to 1.336]
Statistical Analysis 2: Comparison: Tiotropium 5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; Causes of death from MACE were determined by adjudication; Test type: Superiority or Other; p = 0.3263, Regression, Cox; Hazard Ratio (HR) = 1.100, 95% CI 2-sided [0.909 to 1.331]
Statistical Analysis 3: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 5 mcg and Placebo; Causes of death from MACE were determined by adjudication; Test type: Superiority or Other; p = 0.9644, Regression, Cox; Hazard Ratio (HR) = 1.004, 95% CI 2-sided [0.834 to 1.209]

9. Secondary Outcome: Time to Death From Major Adverse Cardiovascular Event (MACE)
Description: The results presented below are number of patients with death from MACE.
Time Frame: Up to 3 years
Population: TS including vital status follow-up, DAS
Measure: Number; unit: Number of deaths from MACE
Arm/Group | Tiotropium 2.5 mcg and Placebo | Tiotropium 5 mcg and Placebo | Tiotropium 18 mcg and Placebo
Number analyzed (Participants) | 5730 | 5711 | 5694
Number of deaths from MACE | 119 | 113 | 101
Statistical Analysis 1: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; Time to death from MACE was analyzed using the full study duration including vital status follow-up; Test type: Superiority or Other; p = 0.2439, Regression, Cox; Hazard Ratio (HR) = 1.171, 95% CI 2-sided [0.898 to 1.526]
Statistical Analysis 2: Comparison: Tiotropium 5 mcg and Placebo vs Tiotropium 18 mcg and Placebo; Time to death from MACE was analyzed using the full study duration including vital status follow-up; Test type: Superiority or Other; p = 0.4413, Regression, Cox; Hazard Ratio (HR) = 1.111, 95% CI 2-sided [0.850 to 1.453]
Statistical Analysis 3: Comparison: Tiotropium 2.5 mcg and Placebo vs Tiotropium 5 mcg and Placebo; Time to death from MACE was analyzed using the full study duration including vital status follow-up; Test type: Superiority or Other; p = 0.6910, Regression, Cox; Hazard Ratio (HR) = 1.054, 95% CI 2-sided [0.814 to 1.363]

ADVERSE EVENTS:
Time Frame: From the first drug intake up to 30 days after administration
Description: Prospectively defined outcome events, serious adverse events, adverse events leading to discontinuation, and investigator-determined drug-related adverse events were required for collection in this trial.
Arm/Group | Tiotropium 2.5 mcg and Placebo | Tiotropium 5 mcg and Placebo | Tiotropium 18 mcg and Placebo
Serious Adverse Events (participants affected / at risk) | 1932/5724 | 1876/5705 | 1928/5687
Other Adverse Events (participants affected / at risk) | 1932/5724 | 1876/5705 | 1928/5687
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium 2.5 mcg and Placebo (N=5724) | Tiotropium 5 mcg and Placebo (N=5705) | Tiotropium 18 mcg and Placebo (N=5687)
Anaemia (Blood and lymphatic system disorders) | 10 | 10 | 13
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 4
Hypercoagulation (Blood and lymphatic system disorders) | 1 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 3 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Pernicious anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 4 | 3 | 9
Acute myocardial infarction (Cardiac disorders) | 21 | 21 | 13
Adams-Stokes syndrome (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 20 | 28 | 22
Angina unstable (Cardiac disorders) | 10 | 19 | 10
Aortic valve disease (Cardiac disorders) | 1 | 0 | 0
Aortic valve disease mixed (Cardiac disorders) | 0 | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 3
Aortic valve stenosis (Cardiac disorders) | 2 | 3 | 3
Arrhythmia (Cardiac disorders) | 5 | 8 | 7
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 41 | 37 | 32
Atrial flutter (Cardiac disorders) | 10 | 6 | 4
Atrial tachycardia (Cardiac disorders) | 2 | 0 | 3
Atrioventricular block (Cardiac disorders) | 3 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 2 | 1 | 2
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 4 | 2 | 2
Bundle branch block left (Cardiac disorders) | 0 | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 12 | 7 | 9
Cardiac asthma (Cardiac disorders) | 1 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 30 | 23 | 24
Cardiac failure acute (Cardiac disorders) | 4 | 4 | 6
Cardiac failure chronic (Cardiac disorders) | 2 | 2 | 3
Cardiac failure congestive (Cardiac disorders) | 26 | 22 | 29
Cardiac valve disease (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 9 | 5 | 8
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 3 | 4 | 3
Cardiomyopathy alcoholic (Cardiac disorders) | 1 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 9 | 11 | 9
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 3 | 1
Cor pulmonale (Cardiac disorders) | 4 | 4 | 6
Cor pulmonale acute (Cardiac disorders) | 1 | 0 | 1
Cor pulmonale chronic (Cardiac disorders) | 3 | 2 | 4
Coronary artery disease (Cardiac disorders) | 18 | 25 | 23
Coronary artery insufficiency (Cardiac disorders) | 2 | 1 | 1
Coronary artery occlusion (Cardiac disorders) | 2 | 2 | 2
Coronary artery stenosis (Cardiac disorders) | 6 | 2 | 3
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 1 | 4
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 2 | 2 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 53 | 45 | 39
Myocardial ischaemia (Cardiac disorders) | 7 | 7 | 11
Palpitations (Cardiac disorders) | 1 | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 1 | 2
Pericarditis (Cardiac disorders) | 1 | 1 | 2
Postinfarction angina (Cardiac disorders) | 0 | 0 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 2 | 2 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 2 | 1
Silent myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 3 | 6
Tachyarrhythmia (Cardiac disorders) | 0 | 2 | 1
Tachycardia (Cardiac disorders) | 3 | 2 | 2
Ventricular arrhythmia (Cardiac disorders) | 0 | 2 | 0
Ventricular dysfunction (Cardiac disorders) | 1 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 3 | 2 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 2 | 3
Alpha-1 anti-trypsin deficiency (Congenital, familial and genetic disorders) | 0 | 0 | 1
Congenital absence of bile ducts (Congenital, familial and genetic disorders) | 1 | 0 | 0
Hamartoma (Congenital, familial and genetic disorders) | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 2 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 6 | 1 | 2
Adrenal mass (Endocrine disorders) | 1 | 0 | 1
Goitre (Endocrine disorders) | 1 | 2 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 2 | 0 | 2
Thyroid mass (Endocrine disorders) | 1 | 0 | 0
Amaurosis (Eye disorders) | 0 | 1 | 0
Amaurosis fugax (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 13 | 10 | 14
Cataract subcapsular (Eye disorders) | 0 | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 1
Lens dislocation (Eye disorders) | 0 | 0 | 1
Macular degeneration (Eye disorders) | 1 | 1 | 0
Open angle glaucoma (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 3 | 2
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1
Retinal infarction (Eye disorders) | 1 | 0 | 0
Strabismus (Eye disorders) | 0 | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 3 | 3
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 13 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 2 | 0 | 1
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 2
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 4 | 0 | 2
Colitis ischaemic (Gastrointestinal disorders) | 1 | 2 | 2
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 1 | 0 | 0
Colonic stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 3 | 4
Crohn's disease (Gastrointestinal disorders) | 3 | 2 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 7
Diverticular perforation (Gastrointestinal disorders) | 1 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 2 | 1 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1 | 0
Duodenal scarring (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 6 | 2 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 2 | 3
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 3 | 2
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 1 | 0
Epiploic appendagitis (Gastrointestinal disorders) | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 3 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 4 | 1 | 4
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 7 | 6 | 4
Gastritis atrophic (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 3 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 2 | 0 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 11 | 12 | 8
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 3 | 3
Gastrooesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 2 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 3 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 3 | 0 | 3
Hiatus hernia (Gastrointestinal disorders) | 2 | 2 | 3
Ileus (Gastrointestinal disorders) | 2 | 3 | 8
Ileus paralytic (Gastrointestinal disorders) | 2 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 10 | 16 | 15
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 3 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 9 | 6 | 7
Intestinal perforation (Gastrointestinal disorders) | 1 | 1 | 1
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 1 | 1
Jejunal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 1 | 1
Large intestine polyp (Gastrointestinal disorders) | 3 | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Lumbar hernia (Gastrointestinal disorders) | 1 | 0 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 1 | 0
Megacolon (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 3 | 2 | 3
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 6
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal food impaction (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 2 | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 9 | 3 | 4
Pancreatitis acute (Gastrointestinal disorders) | 5 | 3 | 4
Pancreatitis chronic (Gastrointestinal disorders) | 4 | 1 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatolithiasis (Gastrointestinal disorders) | 1 | 0 | 0
Papilla of Vater stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Proctocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 5 | 2
Rectal prolapse (Gastrointestinal disorders) | 0 | 1 | 0
Reflux gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Retroperitoneal mass (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 6 | 7 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 2 | 1
Umbilical hernia (Gastrointestinal disorders) | 5 | 1 | 2
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 3 | 3
Volvulus (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 4 | 3 | 3
Adverse drug reaction (General disorders) | 2 | 1 | 3
Asthenia (General disorders) | 8 | 3 | 3
Cardiac death (General disorders) | 1 | 0 | 2
Chest discomfort (General disorders) | 1 | 3 | 3
Chest pain (General disorders) | 4 | 8 | 6
Condition aggravated (General disorders) | 0 | 1 | 0
Cyst (General disorders) | 0 | 0 | 1
Death (General disorders) | 28 | 21 | 13
Device dislocation (General disorders) | 0 | 2 | 0
Device failure (General disorders) | 0 | 0 | 1
Device lead damage (General disorders) | 0 | 0 | 1
Device malfunction (General disorders) | 0 | 0 | 2
Device occlusion (General disorders) | 1 | 0 | 0
Drowning (General disorders) | 0 | 0 | 1
Drug withdrawal syndrome (General disorders) | 1 | 0 | 1
Effusion (General disorders) | 0 | 0 | 1
Exercise tolerance decreased (General disorders) | 0 | 0 | 1
Fibrosis (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 1 | 2 | 1
Hernia (General disorders) | 3 | 3 | 4
Hernia obstructive (General disorders) | 0 | 1 | 0
Hyperthermia (General disorders) | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 1 | 0
Implant site calcification (General disorders) | 0 | 1 | 0
Implant site inflammation (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 1
Mass (General disorders) | 1 | 0 | 0
Multi-organ disorder (General disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 2 | 3 | 7
Necrosis (General disorders) | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 19 | 23 | 22
Oedema (General disorders) | 0 | 1 | 2
Oedema peripheral (General disorders) | 2 | 0 | 5
Polyp (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 3 | 5
Spinal pain (General disorders) | 0 | 0 | 2
Sudden cardiac death (General disorders) | 3 | 9 | 6
Sudden death (General disorders) | 27 | 13 | 18
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0
Ulcer haemorrhage (General disorders) | 1 | 0 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 1 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 3 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 3 | 2 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0
Biliary cyst (Hepatobiliary disorders) | 0 | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 11 | 7 | 6
Cholecystitis acute (Hepatobiliary disorders) | 10 | 2 | 10
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 12 | 12 | 4
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 2
Hepatic congestion (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 0 | 1
Hepatic ischaemia (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 2 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 2 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Amyloidosis (Immune system disorders) | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 2 | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1
Autoimmune disorder (Immune system disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 1
Food allergy (Immune system disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 2 | 1
Abdominal abscess (Infections and infestations) | 0 | 1 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 2 | 0
Abscess intestinal (Infections and infestations) | 1 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 3
Abscess neck (Infections and infestations) | 1 | 0 | 0
Acinetobacter infection (Infections and infestations) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 2
Amoebic dysentery (Infections and infestations) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 1 | 0
Anal infection (Infections and infestations) | 0 | 0 | 1
Appendiceal abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 7 | 6 | 7
Appendicitis perforated (Infections and infestations) | 3 | 2 | 2
Arthritis bacterial (Infections and infestations) | 2 | 0 | 0
Arthritis infective (Infections and infestations) | 2 | 0 | 1
Atypical mycobacterial infection (Infections and infestations) | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Bacterial toxaemia (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 16 | 9 | 11
Bronchitis bacterial (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 4 | 3 | 4
Bursitis infective (Infections and infestations) | 0 | 2 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 1
Campylobacter infection (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 6 | 14 | 14
Cellulitis of male external genital organ (Infections and infestations) | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0
Chronic hepatitis C (Infections and infestations) | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 3
Clostridium colitis (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 3 | 2
Clostridium difficile infection (Infections and infestations) | 3 | 2 | 0
Colon gangrene (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 2 | 3 | 4
Dengue fever (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 1 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 9 | 6 | 6
Ear infection (Infections and infestations) | 1 | 0 | 0
Eczema infected (Infections and infestations) | 0 | 1 | 0
Empyema (Infections and infestations) | 0 | 1 | 3
Endocarditis (Infections and infestations) | 0 | 3 | 3
Endophthalmitis (Infections and infestations) | 1 | 0 | 1
Enterobacter pneumonia (Infections and infestations) | 0 | 1 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 1
Enterocolitis viral (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 2 | 2 | 3
Eye infection (Infections and infestations) | 0 | 1 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 2 | 0 | 1
Gallbladder empyema (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 2 | 1
Gastritis viral (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 11 | 5 | 8
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 1
Gastroenteritis clostridial (Infections and infestations) | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 1 | 0
Groin abscess (Infections and infestations) | 2 | 0 | 0
Groin infection (Infections and infestations) | 0 | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 0 | 0
Haematoma infection (Infections and infestations) | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 1
Hepatic cyst infection (Infections and infestations) | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 2 | 0 | 0
Hepatitis viral (Infections and infestations) | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 3 | 2 | 2
Herpes zoster ophthalmic (Infections and infestations) | 0 | 0 | 1
Herpes zoster oticus (Infections and infestations) | 0 | 0 | 1
Implant site infection (Infections and infestations) | 1 | 1 | 0
Incision site infection (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 2 | 4
Infectious pleural effusion (Infections and infestations) | 1 | 2 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 16 | 8 | 8
Influenza (Infections and infestations) | 4 | 6 | 2
Intervertebral discitis (Infections and infestations) | 2 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 1
Liver abscess (Infections and infestations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 16 | 15 | 12
Localised infection (Infections and infestations) | 2 | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 2
Lung abscess (Infections and infestations) | 2 | 2 | 2
Lung infection (Infections and infestations) | 0 | 1 | 3
Lyme disease (Infections and infestations) | 0 | 1 | 2
Mastitis (Infections and infestations) | 0 | 0 | 1
Measles (Infections and infestations) | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0
Nosocomial infection (Infections and infestations) | 0 | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 2 | 1 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 3 | 1 | 1
Otitis media (Infections and infestations) | 0 | 1 | 1
Pelvic abscess (Infections and infestations) | 0 | 0 | 2
Perineal abscess (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 4 | 2 | 1
Pertussis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumocystis jiroveci infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 339 | 344 | 340
Pneumonia bacterial (Infections and infestations) | 4 | 1 | 1
Pneumonia influenzal (Infections and infestations) | 2 | 0 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0 | 0
Pneumonia necrotising (Infections and infestations) | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1
Pneumonia pseudomonas aeruginosa (Infections and infestations) | 1 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 1 | 2
Pneumonia streptococcal (Infections and infestations) | 0 | 1 | 1
Pneumonia viral (Infections and infestations) | 1 | 0 | 0
Postoperative abscess (Infections and infestations) | 0 | 0 | 2
Postoperative wound infection (Infections and infestations) | 0 | 1 | 3
Pseudomembranous colitis (Infections and infestations) | 0 | 2 | 0
Pseudomonas bronchitis (Infections and infestations) | 0 | 1 | 0
Psoas abscess (Infections and infestations) | 0 | 1 | 0
Pulmonary tuberculoma (Infections and infestations) | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 5
Purulence (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 6 | 6 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 1 | 2
Pyoderma (Infections and infestations) | 1 | 0 | 0
Pyonephrosis (Infections and infestations) | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 3 | 7 | 3
Scrotal abscess (Infections and infestations) | 1 | 2 | 0
Sepsis (Infections and infestations) | 18 | 22 | 16
Sepsis syndrome (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 6 | 6 | 12
Serratia infection (Infections and infestations) | 0 | 1 | 0
Sialoadenitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 0
Skin infection (Infections and infestations) | 1 | 1 | 1
Soft tissue infection (Infections and infestations) | 1 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 2 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1 | 2
Tracheobronchitis (Infections and infestations) | 0 | 1 | 1
Tuberculosis (Infections and infestations) | 2 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 3
Urethral abscess (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 9 | 22 | 6
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 7 | 2 | 4
Vestibular neuronitis (Infections and infestations) | 1 | 1 | 1
Viral diarrhoea (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 1 | 0
Wound infection (Infections and infestations) | 2 | 3 | 3
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 1 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1
Arterial restenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 1 | 1
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 1 | 4
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 | 1 | 1
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 3 | 2
Fall (Injury, poisoning and procedural complications) | 8 | 19 | 4
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 3 | 5
Femur fracture (Injury, poisoning and procedural complications) | 5 | 5 | 4
Fibula fracture (Injury, poisoning and procedural complications) | 3 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 3 | 1
Foreign body (Injury, poisoning and procedural complications) | 3 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 11 | 5 | 11
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 4 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 3 | 2 | 1
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Injury corneal (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 3 | 2 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 5 | 0 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2 | 1
Open fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 3 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1
Pneumoconiosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 2 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 2
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 4 | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 10 | 9 | 5
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 3 | 5
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin graft failure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 4 | 2 | 4
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 6 | 1 | 2
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Splinter (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 2 | 5
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 3 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 2 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 5 | 2 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 2 | 4
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 6 | 3 | 0
Urethral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 | 0 | 2
Wound (Injury, poisoning and procedural complications) | 1 | 1 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 1 | 4
Angiogram (Investigations) | 1 | 0 | 0
Arteriogram coronary normal (Investigations) | 0 | 1 | 0
Arthroscopy (Investigations) | 0 | 0 | 1
Biopsy lung (Investigations) | 1 | 1 | 0
Biopsy vocal cord normal (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 1
Catheterisation cardiac (Investigations) | 2 | 1 | 2
Chest X-ray abnormal (Investigations) | 1 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 1 | 0
Full blood count decreased (Investigations) | 0 | 0 | 1
International normalised ratio abnormal (Investigations) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0
Investigation (Investigations) | 0 | 0 | 1
Laparoscopy (Investigations) | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 1
Prostatic specific antigen increased (Investigations) | 1 | 0 | 0
Troponin I increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 4 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 8 | 8 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 4 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1 | 2
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 0 | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 4
Feeding disorder (Metabolism and nutrition disorders) | 0 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 4 | 5
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 2 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 5 | 8 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 3 | 6
Bone infarction (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursa disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Chondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 10 | 6 | 10
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 | 12 | 23
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 6 | 1 | 2
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 4 | 6
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Acral lentiginous melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3
B-cell unclassifiable lymphoma low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 | 26 | 15
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign neoplasm of urethra (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 10 | 4
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 4
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 8 | 4
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 7 | 4
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 4 | 10
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3 | 4
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Large cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 9 | 6
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 7 | 9
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 7 | 5
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 52 | 60 | 48
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 4
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant splenic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 0 | 2
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3 | 3
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Metastases to muscle (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Metastases to retroperitoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1
Metastases to spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Nasal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Nasopharyngeal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Nasopharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5 | 5
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-small cell lung cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Oropharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6 | 7
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 3
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 | 17 | 14
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 3
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5 | 4
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 12 | 19
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6 | 6
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 2
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5 | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Urinary tract carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vascular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1
Brain hypoxia (Nervous system disorders) | 0 | 0 | 1
Brain injury (Nervous system disorders) | 0 | 1 | 3
Brain oedema (Nervous system disorders) | 1 | 0 | 1
Brain stem infarction (Nervous system disorders) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 4 | 8 | 7
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 2
Cauda equina syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebellar ataxia (Nervous system disorders) | 1 | 0 | 0
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 1 | 0
Cerebral artery embolism (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 4 | 4 | 2
Cerebral infarction (Nervous system disorders) | 2 | 2 | 2
Cerebral ischaemia (Nervous system disorders) | 2 | 1 | 0
Cerebral thrombosis (Nervous system disorders) | 0 | 0 | 1
Cerebrosclerosis (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 35 | 38 | 35
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 1
Cervical myelopathy (Nervous system disorders) | 1 | 0 | 0
Coma (Nervous system disorders) | 1 | 0 | 0
Complicated migraine (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 3 | 2 | 5
Dementia (Nervous system disorders) | 1 | 4 | 1
Dementia Alzheimer's type (Nervous system disorders) | 2 | 0 | 0
Demyelinating polyneuropathy (Nervous system disorders) | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 5 | 3
Dysarthria (Nervous system disorders) | 1 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1 | 0
Encephalitis (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 2 | 4 | 3
Facial spasm (Nervous system disorders) | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 1
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 3 | 0
Headache (Nervous system disorders) | 2 | 3 | 3
Hemiplegia (Nervous system disorders) | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 1 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0 | 0
Hypertonia (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2 | 1 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 3 | 1 | 0
Intracranial haematoma (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 5 | 3 | 7
Lacunar infarction (Nervous system disorders) | 1 | 1 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 2 | 1 | 0
Motor dysfunction (Nervous system disorders) | 0 | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 1 | 0
Peripheral nerve lesion (Nervous system disorders) | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 2 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 2
Quadriplegia (Nervous system disorders) | 0 | 1 | 0
Radial nerve palsy (Nervous system disorders) | 0 | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 3 | 2 | 2
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Spinal cord infarction (Nervous system disorders) | 0 | 0 | 1
Spinal cord ischaemia (Nervous system disorders) | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 3 | 0 | 2
Syncope (Nervous system disorders) | 14 | 17 | 15
Tension headache (Nervous system disorders) | 0 | 1 | 0
Tongue biting (Nervous system disorders) | 0 | 0 | 1
Tonic convulsion (Nervous system disorders) | 0 | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 18 | 23 | 14
Tremor (Nervous system disorders) | 1 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0
Ulnar tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 1 | 0
Vascular dementia (Nervous system disorders) | 1 | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 0 | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 1 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 1
Alcoholic psychosis (Psychiatric disorders) | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 2 | 3 | 0
Anxiety (Psychiatric disorders) | 2 | 5 | 2
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 2 | 2
Confusional state (Psychiatric disorders) | 1 | 0 | 3
Delirium (Psychiatric disorders) | 3 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 7 | 7 | 5
Disorientation (Psychiatric disorders) | 0 | 1 | 0
Drug abuse (Psychiatric disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0
Mania (Psychiatric disorders) | 0 | 2 | 0
Mental disorder (Psychiatric disorders) | 1 | 2 | 0
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 2 | 2
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 1
Stress (Psychiatric disorders) | 1 | 1 | 0
Substance abuse (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 2 | 2
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0 | 0
Bladder cyst (Renal and urinary disorders) | 1 | 0 | 0
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 0 | 1
Bladder perforation (Renal and urinary disorders) | 1 | 0 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 3 | 0
Calculus urethral (Renal and urinary disorders) | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 4
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 3 | 9 | 4
Hydronephrosis (Renal and urinary disorders) | 0 | 3 | 0
Ketonuria (Renal and urinary disorders) | 1 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 4 | 8 | 4
Nephropathy (Renal and urinary disorders) | 0 | 2 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 0 | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0
Postrenal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 3
Renal failure (Renal and urinary disorders) | 9 | 8 | 5
Renal failure acute (Renal and urinary disorders) | 17 | 14 | 24
Renal failure chronic (Renal and urinary disorders) | 2 | 2 | 2
Renal impairment (Renal and urinary disorders) | 2 | 1 | 1
Renal infarct (Renal and urinary disorders) | 0 | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 2
Urethral stenosis (Renal and urinary disorders) | 0 | 2 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 5 | 9 | 9
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Acquired phimosis (Reproductive system and breast disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 8 | 14 | 4
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 2 | 1 | 2
Ovarian mass (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatic dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 5 | 2 | 1
Rectocele (Reproductive system and breast disorders) | 1 | 0 | 1
Spermatic cord inflammation (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 30 | 32 | 28
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 7
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 895 | 868 | 851
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 17 | 21
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 13
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 8
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Laryngeal leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngeal polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural calcification (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 10
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 25 | 25 | 21
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 28 | 28 | 24
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 10
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 42 | 40 | 35
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Peau d'orange (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Abstains from alcohol (Social circumstances) | 0 | 1 | 0
Cardiac assistance device user (Social circumstances) | 1 | 0 | 0
Angioplasty (Surgical and medical procedures) | 0 | 0 | 2
Aortic valve repair (Surgical and medical procedures) | 0 | 1 | 0
Aortic valve replacement (Surgical and medical procedures) | 1 | 0 | 1
Appendicectomy (Surgical and medical procedures) | 0 | 1 | 0
Arterial repair (Surgical and medical procedures) | 0 | 0 | 1
Arterial stent insertion (Surgical and medical procedures) | 1 | 0 | 1
Bladder neoplasm surgery (Surgical and medical procedures) | 1 | 0 | 0
Bladder operation (Surgical and medical procedures) | 0 | 0 | 1
Bone graft (Surgical and medical procedures) | 0 | 0 | 1
Bone operation (Surgical and medical procedures) | 0 | 0 | 1
Cardiac ablation (Surgical and medical procedures) | 0 | 1 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 1 | 2
Cardiac pacemaker removal (Surgical and medical procedures) | 1 | 0 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 | 2 | 1
Central venous catheterisation (Surgical and medical procedures) | 1 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 5 | 5 | 1
Cholecystostomy (Surgical and medical procedures) | 1 | 0 | 0
Colon operation (Surgical and medical procedures) | 0 | 1 | 0
Colostomy (Surgical and medical procedures) | 1 | 0 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 2 | 0 | 1
Coronary artery bypass (Surgical and medical procedures) | 1 | 2 | 2
Coronary endarterectomy (Surgical and medical procedures) | 0 | 0 | 1
Coronary revascularisation (Surgical and medical procedures) | 1 | 0 | 0
Dental implantation (Surgical and medical procedures) | 0 | 0 | 1
Ear operation (Surgical and medical procedures) | 0 | 0 | 1
Elective surgery (Surgical and medical procedures) | 1 | 0 | 0
Endobronchial valve implantation (Surgical and medical procedures) | 1 | 1 | 1
Frontal sinus operation (Surgical and medical procedures) | 0 | 0 | 1
Gallbladder operation (Surgical and medical procedures) | 1 | 0 | 0
Gastroenterostomy (Surgical and medical procedures) | 1 | 0 | 0
Haemorrhoid operation (Surgical and medical procedures) | 0 | 2 | 0
Heart valve operation (Surgical and medical procedures) | 0 | 0 | 1
Heart valve replacement (Surgical and medical procedures) | 0 | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 2 | 4
Hip surgery (Surgical and medical procedures) | 0 | 2 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 1 | 0
Hysterectomy (Surgical and medical procedures) | 2 | 0 | 0
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 1 | 0 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 0 | 2 | 1
Implantable defibrillator replacement (Surgical and medical procedures) | 0 | 0 | 1
Inguinal hernia repair (Surgical and medical procedures) | 2 | 1 | 0
Intervertebral disc operation (Surgical and medical procedures) | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 3 | 6 | 4
Large intestine anastomosis (Surgical and medical procedures) | 0 | 0 | 1
Leg amputation (Surgical and medical procedures) | 0 | 0 | 1
Limb operation (Surgical and medical procedures) | 1 | 2 | 0
Lung transplant (Surgical and medical procedures) | 0 | 0 | 1
Lung volume reduction surgery (Surgical and medical procedures) | 1 | 0 | 1
Mechanical ventilation (Surgical and medical procedures) | 1 | 1 | 1
Medical device change (Surgical and medical procedures) | 1 | 0 | 0
Medical device removal (Surgical and medical procedures) | 0 | 0 | 1
Nasal septal operation (Surgical and medical procedures) | 1 | 0 | 0
Obesity surgery (Surgical and medical procedures) | 0 | 0 | 1
Partial lung resection (Surgical and medical procedures) | 0 | 0 | 1
Peripheral artery bypass (Surgical and medical procedures) | 1 | 0 | 0
Polypectomy (Surgical and medical procedures) | 0 | 1 | 0
Prophylaxis (Surgical and medical procedures) | 0 | 0 | 1
Prostatectomy (Surgical and medical procedures) | 2 | 1 | 0
Prostatic operation (Surgical and medical procedures) | 0 | 3 | 0
Prosthesis implantation (Surgical and medical procedures) | 0 | 1 | 0
Pulmonary valve replacement (Surgical and medical procedures) | 0 | 0 | 1
Rehabilitation therapy (Surgical and medical procedures) | 1 | 0 | 0
Respiratory therapy (Surgical and medical procedures) | 1 | 0 | 0
Rotator cuff repair (Surgical and medical procedures) | 0 | 1 | 0
Salpingo-oophorectomy (Surgical and medical procedures) | 0 | 0 | 1
Shoulder arthroplasty (Surgical and medical procedures) | 2 | 1 | 0
Shoulder operation (Surgical and medical procedures) | 1 | 0 | 0
Skin operation (Surgical and medical procedures) | 0 | 1 | 0
Spinal fusion surgery (Surgical and medical procedures) | 0 | 1 | 0
Spinal laminectomy (Surgical and medical procedures) | 0 | 2 | 1
Spinal operation (Surgical and medical procedures) | 1 | 0 | 0
Stem cell transplant (Surgical and medical procedures) | 0 | 0 | 1
Stent placement (Surgical and medical procedures) | 0 | 0 | 2
Surgery (Surgical and medical procedures) | 0 | 1 | 1
Thyroidectomy (Surgical and medical procedures) | 0 | 2 | 0
Transurethral bladder resection (Surgical and medical procedures) | 0 | 0 | 1
Transurethral prostatectomy (Surgical and medical procedures) | 2 | 1 | 2
Urethral operation (Surgical and medical procedures) | 0 | 0 | 1
Urethrotomy (Surgical and medical procedures) | 0 | 1 | 0
Vaginoplasty (Surgical and medical procedures) | 1 | 0 | 0
Vascular graft (Surgical and medical procedures) | 1 | 0 | 1
Vascular stent insertion (Surgical and medical procedures) | 0 | 1 | 1
Accelerated hypertension (Vascular disorders) | 1 | 0 | 0
Aneurysm (Vascular disorders) | 0 | 4 | 0
Aneurysm ruptured (Vascular disorders) | 2 | 0 | 0
Aortic aneurysm (Vascular disorders) | 8 | 15 | 12
Aortic aneurysm rupture (Vascular disorders) | 2 | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0 | 1
Aortic occlusion (Vascular disorders) | 0 | 1 | 0
Aortic rupture (Vascular disorders) | 2 | 0 | 0
Aortic stenosis (Vascular disorders) | 2 | 4 | 1
Arterial disorder (Vascular disorders) | 1 | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1 | 0
Arterial occlusive disease (Vascular disorders) | 2 | 3 | 2
Arterial stenosis (Vascular disorders) | 0 | 2 | 0
Arterial thrombosis (Vascular disorders) | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 5 | 6 | 4
Arteritis (Vascular disorders) | 0 | 1 | 0
Bleeding varicose vein (Vascular disorders) | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 4 | 2 | 1
Deep vein thrombosis (Vascular disorders) | 5 | 11 | 6
Embolism (Vascular disorders) | 1 | 0 | 0
Extremity necrosis (Vascular disorders) | 1 | 1 | 1
Femoral artery occlusion (Vascular disorders) | 1 | 2 | 1
Haematoma (Vascular disorders) | 0 | 1 | 4
Haemorrhage (Vascular disorders) | 2 | 0 | 2
Hypertension (Vascular disorders) | 8 | 8 | 12
Hypertensive crisis (Vascular disorders) | 4 | 2 | 1
Hypotension (Vascular disorders) | 0 | 6 | 9
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 2
Iliac artery occlusion (Vascular disorders) | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 4 | 2 | 3
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1
Leriche syndrome (Vascular disorders) | 0 | 1 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 4
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 7 | 8 | 10
Peripheral artery aneurysm (Vascular disorders) | 0 | 2 | 0
Peripheral artery stenosis (Vascular disorders) | 4 | 3 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 2 | 1
Peripheral ischaemia (Vascular disorders) | 4 | 5 | 3
Peripheral vascular disorder (Vascular disorders) | 4 | 2 | 1
Post thrombotic syndrome (Vascular disorders) | 1 | 1 | 0
Shock (Vascular disorders) | 2 | 1 | 1
Shock haemorrhagic (Vascular disorders) | 2 | 0 | 0
Steal syndrome (Vascular disorders) | 0 | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 1
Thrombosis (Vascular disorders) | 4 | 0 | 3
Varicose vein (Vascular disorders) | 2 | 0 | 0
Vascular occlusion (Vascular disorders) | 2 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 2
Vasodilatation (Vascular disorders) | 0 | 1 | 1
Venous insufficiency (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 2 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium 2.5 mcg and Placebo (N=5724) | Tiotropium 5 mcg and Placebo (N=5705) | Tiotropium 18 mcg and Placebo (N=5687)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1932 | 1876 | 1928

LIMITATIONS AND CAVEATS:
Prospectively defined outcome events, serious adverse events, adverse events leading to discontinuation, and investigator-determined drug-related adverse events were required for collection in this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.